## Johnson & Johnson Vision Care, Inc.

## Clinical Study Protocol

Evaluation of a Toric Multifocal Contact Lens Manufactured in Etafilcon Material in a Low ADD Hyperopic Population

Protocol CR-6278

Version: 1.0

Date: 12 July 2018.

Investigational Products: JJV Investigational Toric Multifocal Contact Lenses manufactured in etafilcon A material

Key Words: Presbyopia, Multifocal, Astigmatism, Daily Disposable, Dispensing, Etafilcon A

### Statement of Compliance to protocol, GCP and applicable regulatory guidelines:

This trial will be conducted in compliance with the protocol, ISO 14155,<sup>1</sup> the International Conference on Harmonization Good Clinical Practice E6 (ICH-GCP),<sup>2</sup> the Declaration of Helsinki,<sup>3</sup> and all applicable regulatory requirements.

#### **Confidentiality Statement:**

This document contains confidential information, which should not be copied, referred to, released or published without written approval from Johnson & Johnson Vision Care, Inc. The information may not be disclosed to others except to the extent necessary to obtain Institutional Review Board/Independent Ethics Committee approval and informed consent, or as required by International, Federal and State Laws, as applicable. Persons to whom this information is disclosed must be informed that this information is privileged and confidential and that it should not be further disclosed without the written permission of Johnson & Johnson Vision Care, Inc. Any supplemental information that may be added to this document is also confidential and proprietary to Johnson & Johnson Vision Care, Inc. and must be kept in confidence in the same manner as the contents of this document.

# TABLE OF CONTENTS

| PROT | OCOL TITLE, NUMBER, VERSION | 6 |
|---|---|---|
| SPON | SOR NAME AND ADDRESS | 6 |
| MEDI | CAL MONITOR | 6 |
| AUTH | IORIZED SIGNATURES | 7 |
| CHAN | NGE HISTORY | 8 |
| SYNO | PSIS | 9 |
| COMN | MONLY USED ABBREVIATIONS AND DEFINITIONS OF TERMS | 13 |
| 1. | INTRODUCTION AND BACKGROUND | 15 |
| 1.1. | Name and Descriptions of Investigational Products | 15 |
| 1.2. | Intended Use of Investigational Products | 15 |
| 1.3. | Summary of Findings from Nonclinical Studies | 15 |
| 1.4. | Summary of Known Risks and Benefits to Human Subjects | 15 |
| _ | .5. Relevant Literature References and Prior Clinical Data Relevant to Propos | |
| | y | |
| 2. | STUDY OBJECTIVES, ENDPOINTS AND HYPOTHESES | |
| 2.1. | Objectives | |
| 2.2. | Endpoints | |
| 2.3. | Hypotheses | |
| 3. | TARGETED STUDY POPULATION | |
| 3.1. | General Characteristics | |
| 3.2. | Inclusion Criteria | |
| 3.3.<br>3.4. | Exclusion Criteria | |
| 3.4.<br>4. | STUDY DESIGN AND RATIONALE | |
| 4.1. | Description of Study Design | |
| 4.2. | Study Design Rationale | |
| 4.2. | Enrollment Target and Study Duration | |
| 5. | TEST ARTICLE ALLOCATION AND MASKING | |
| <i>5</i> . 5.1. | Test Article Allocation | |
| 5.2. | Masking | |
| 5.3. | Procedures for Maintaining and Breaking the Masking | |
| 6. | STUDY INTERVENTION | |

| 6.1. | Identity of Test Articles | . 21 |
|---|---|---|
| 6.2. | Ancillary Supplies/Products | . 22 |
| 6.3. | Administration of Test Articles | . 22 |
| 6.4. | Packaging and Labeling | . 22 |
| 6.5. | Storage Conditions | . 23 |
| 6.6. | Collection and Storage of Samples | . 23 |
| 6.7. | Accountability of Test Articles | . 23 |
| 7. | STUDY EVALUATIONS | . 24 |
| 7.1. | Time and Event Schedule | . 24 |
| 7.2. | Detailed Study Procedures | . 27 |
| VI | SIT 1 | . 27 |
| VI | SIT 2 | . 35 |
| VI | SIT 3 | . 42 |
| FI | NAL EVALUATION | . 45 |
| 7.3. | Unscheduled Visits | . 45 |
| 7.4. | Laboratory Procedures | . 47 |
| 8. | SUBJECTS COMPLETION/WITHDRAWAL | . 47 |
| 8.1. | Completion Criteria | . 47 |
| 8.2. | Withdrawal/Discontinuation from the Study | . 47 |
| 9. | PRE-STUDY AND CONCOMITANT INTERVENTION/MEDICATION | . 48 |
| 10. | DEVIATIONS FROM THE PROTOCOL | |
| 11. | STUDY TERMINATION | . 48 |
| 12. | PROCEDURE FOR HANDLING PRODUCT QUALITY COMPLAINTS | |
| 13. | ADVERSE EVENTS | . 50 |
| 13.1. | Definitions and Classifications | . 50 |
| 13.2. | Assessing Adverse Events | . 53 |
| 13 | .2.1. Causality Assessment | . 53 |
| 13 | .2.2. Severity Assessment | . 53 |
| 13.3. | Documentation and Follow-Up of Adverse Events | . 54 |
| 13.4. | Reporting Adverse Events | . 55 |
| 13 | .4.1. Reporting Adverse Events to Sponsor | . 55 |
| 13 | .4.2. Reporting Adverse Events to the Responsible IEC/IRB and Health Authorities | |
| 13 | .4.3. Event of Special Interest | . 56 |
| 13.5 | Reporting of Pregnancy | . 56 |

| 14. | STATISTICAL METHODS | 56 |
|---|---|---|
| 14.1. | General Considerations | 56 |
| 14.2. | Sample Size Justification. | 57 |
| 14.3. | Analysis Populations | 58 |
| 14.4. | Level of Statistical Significance | 58 |
| 14.5. | Primary Analysis | 58 |
| 14.6. | Secondary Analysis | 59 |
| 14.7. | Other Exploratory Analyses | 59 |
| 14.8. | Interim Analysis | 59 |
| 14.9. | Procedure for Handling Missing Data and Drop-Outs | 59 |
| 14.10. | Procedure for Reporting Deviations from Statistical Plan | 59 |
| 15. | DATA HANDLING AND RECORD KEEPING/ARCHIVING | 59 |
| 15.1. | Electronic Case Report Form/Data Collection | 59 |
| 15.2. | Subject Record | 60 |
| 16. | DATA MANAGEMENT | 60 |
| 16.1. | Access to Source Data/Document | 60 |
| 16.2. | Confidentiality of Information | 61 |
| 16.3. | Data Quality Assurance | 61 |
| 17. | MONITORING | 61 |
| 18. | ETHICAL AND REGULATORY ASPECTS | 62 |
| 18.1. | Study-Specific Design Considerations | 62 |
| 18.2. | Investigator Responsibility | 62 |
| 18.3. | Independent Ethics Committee or Institutional Review Board (IEC/IRB) | 62 |
| 18.4. | Informed Consent | 63 |
| 18.5. | Privacy of Personal Data | 64 |
| 19. | STUDY RECORD RETENTION | 65 |
| 20. | FINANCIAL CONSIDERATIONS | 65 |
| 21. | PUBLICATION | 66 |
| 22. | REFERENCES | 66 |
| APPEN] | DIX A: PATIENT REPORTED OUTCOMES (STUDY QUESTIONNAIRES) | 67 |
| APPEN | DIX B: PATIENT INSTRUCTION GUIDE | 84 |
| APPEN] | DIX C: PACKAGE INSERT (APPROVED PRODUCT) | 85 |
| APPEN] | DIX D: PRESBYOPIC SYMPTOMS QUESTIONNAIRE | 86 |
| APPEN | DIX E: OCULAR DOMINANCE | 87 |

| APPENDIX F: Test LENS FITTING GUIDE | 88 |
|----------------------------------------------------------|--------|
| APPENDIX G: BINOCULAR OVER REFRACTION | 90 |
| APPENDIX H: | 91 |
| , LIMBAL & CONJUNCTIVAL (BULBAR) REDNESS | 92 |
| , EXPANDED SODIUM FLUORESCEIN CORNEAL STAINING | 100 |
| , DETERMINATION OF NEAR ADD | 105 |
| , NEAR logMAR VISUAL ACUITY MEASUREMENT PROCEDURE | 113 |
| , LENS FITTING CHARACTERISTICS | 116 |
| , SUBJECT REPORTED OCULAR SYMPTOMS | 123 |
| , DETERMINATION OF DISTANCE SPHEROCYLINDRICAL REFRACTION | )NS125 |
| , BIOMICROSCOPY SCALE | 132 |
| , KERATOMETRY | 138 |
| , DISTANCE AND NEAR VISUAL ACUITY EVALUATION | 140 |
| , TORIC FIT EVALUATION | 145 |
| , ETDRS DISTANCE VISUAL ACUITY MEASURMENT PROCEDURE | 149 |
| , LENS INSERTION AND REMOVAL | 153 |
| , VISUAL ACUITY CHART LUMINANCE AND ROOM ILLUMIN | |
| PROTOCOL COMPLIANCE INVESTIGATOR(S) SIGNATURE PAGE | 161 |
| TABLE OF CONTENTS Figure 1: Study Flowchart | 12 |
| TABLE OF CONTENTS | |
| Table 1: Test Articles | 21 |
| Table 2: Ancillary Supplies | |
| Table 3: Time and Events | 24 |

#### PROTOCOL TITLE, NUMBER, VERSION

Title: Evaluation of a Toric Multifocal Contact Lens Manufactured in Etafilcon Material in a Low

ADD Hyperopic Population Protocol Number: CR-6278

Version: 1.0

Date: 12 July 2018

#### SPONSOR NAME AND ADDRESS

Johnson & Johnson Vision Care (JJVC) 7500 Centurion Parkway Jacksonville, FL 32256

#### MEDICAL MONITOR



The Medical Monitor must be notified by the clinical institution/site by e-mail, fax, or telephone within 24 hours of learning of a Serious Adverse Event. The Medical Monitor may be contacted during business hours for adverse event questions. General study related questions should be directed towards your assigned clinical research associate.

The Medical Monitoring Plan is maintained as a separate document and included in the Trial Master File.

#### AUTHORIZED SIGNATURES

The signature below constitutes the approval of this protocol and the attachments, and provides the necessary assurances that this trial will be conducted according to all stipulations of the protocol, including all statements regarding confidentiality, and according to local legal and regulatory requirements and applicable U.S. federal regulations, ICH guidelines, ISO 14155, and the Declaration of Helsinki.

| Author | See Electronic Signature Report | DATE |
|--------------------------------|---------------------------------|------|
| Clinical Operations<br>Manager | See Electronic Signature Report | DATE |
| Biostatistician | See Electronic Signature Report | DATE |
| Data Management | See Electronic Signature Report | DATE |
| Reviewer | Fellow Review Not Required | DATE |
| Approver | See Electronic Signature Report | DATE |

## **CHANGE HISTORY**

| Version | Originator | Description of Change(s) and Section<br>Number(s) Affected | Date |
|---|---|---|---|
| 1.0 | | Original Protocol | 12-Jul-2018 |

## **SYNOPSIS**

| Protocol Title Evaluation of a Toric Multifocal Contact Lens Manufactured in Etafilcon Material in a Low ADD Hyperopic Population Sponsor JJVC, 7500 Centurion Parkway, Jacksonville, FL 32256 Clinical Phase Development phase, Phase 2 Trial Registration This study will be registered on ClinicalTrials.gov. Investigational Product: JJVC Investigational Toric Multifocal Contact Lens manufactured in etafilcon A material. Wear and Replacement Schedules Wear Schedule: The lenses will be used on a daily disposable basis. Replacement Schedule: The lenses will be replaced after a day of wear. Objectives Primary Objective(s) The primary Objectives of this study are an evaluation of the clinical performance of logMAR visual acuity and subjective visual response. Study Endpoints Primary endpoints: logMAR visual acuity, and subjective visual response. Study Design The study is a bilateral, single masked, single-arm, 3-visit dispensing study. There will be one study treatment, with the subject being in the treatment for approximately 12-16 days. A total of approximately 36 cligible subjects will be targeted to complete the study (low Add hyperopes only). The subjects will be fit in the study lens and wear the study lenses for 6-8 days. The primary endpoints of this study are logMAR visual acuity and subjective visual response. See the flow chart at the end of the synopsis table for the schematic of the study visits and procedures of main observations (Figure 1). Sample Size A total of approximately 40 eligible subjects will be enrolled with 36 subjects targeted to complete. The study will last approximately 2 months. Healthy male and female volunteers with presbyopia will be screened as per criteria outlined below. All volunteers will have baseline measurements taken to ensure eligibility. The baseline procedures will occur after inform consent has been obtained. For a detailed list of procedures see the time and events schedule listed below. Eligibility Criteria | | |
|---|---|---|
| Sponsor JJVC, 7500 Centurion Parkway, Jacksonville, FL 32256 | Protocol Title | |
| Development phase Development phase Trial Registration This study will be registered on Clinical Trials.gov. | | |
| Trial Registration Test Article(s) Investigational Product: JIVC Investigational Toric Multifocal Contact Lens manufactured in etafilcon A material. Wear and Replacement Schedules Wear Schedule: The lenses will be used on a daily disposable basis. Replacement Schedule: The lenses will be replaced after a day of wear. Objectives Primary Objective(s) The primary objectives of this study are an evaluation of the clinical performance of logMAR visual acuity and subjective visual response. Study Endpoints Primary endpoints: logMAR visual acuity, and subjective visual response. Study Design The study is a bilateral, single masked, single-arm, 3-visit dispensing study. There will be one study treatment, with the subject being in the treatment for approximately 12-16 days. A total of approximately 36 eligible subjects will be targeted to complete the study (low Add hyperopes only). The subjects will be fit in the study lens and wear the optimized pair for 6-8 days. The primary endpoints of this study are logMAR visual acuity and subjective visual response. See the flow chart at the end of the synopsis table for the schematic of the study visits and procedures of main observations (Figure 1). Sample Size A total of approximately 40 eligible subjects will be enrolled with 36 subjects targeted to complete. Study Duration The study will last approximately 2 months. Healthy male and female volunteers with presbyopia will be screened as per criteria outlined below. All volunteers will have baseline measurements taken to ensure eligibility. The baseline procedures will occur after inform consent has been obtained. For a detailed list of procedures see the time and events schedule listed below. Eligibility Criteria | - | • |
| Test Article(s) Investigational Product: JJVC Investigational Toric Multifocal Contact Lens manufactured in etafilcon A material. Wear and Replacement Schedules Wear Schedule: The lenses will be used on a daily disposable basis. Replacement Schedule: The lenses will be replaced after a day of wear. Objectives Primary Objective(s) The primary objectives of this study are an evaluation of the clinical performance of logMAR visual acuity and subjective visual response. Study Endpoints Primary endpoints: logMAR visual acuity, and subjective visual response. Study Design The study is a bilateral, single masked, single-arm, 3-visit dispensing study. There will be one study treatment, with the subject being in the treatment for approximately 12-16 days. A total of approximately 36 eligible subjects will be targeted to complete the study (low Add hyperopes only). The subjects will be fit in the study lens and wear the study lenses for 6-8 days. The primary endpoints of this study are logMAR visual acuity and subjective visual response. See the flow chart at the end of the synopsis table for the schematic of the study visits and procedures of main observations (Figure 1). Sample Size A total of approximately 40 eligible subjects will be enrolled with 36 subjects targeted to complete. Study Duration The study will last approximately 2 months. Healthy male and female volunteers with presbyopia will be screened as per criteria outlined below. All volunteers will have baseline measurements taken to ensure eligibility. The baseline procedures will occur after inform consent has been obtained. For a detailed list of procedures see the time and events schedule listed below. Eligibility Criteria | | |
| Contact Lens manufactured in etafilcon A material. | | |
| Schedules basis. Replacement Schedule: The lenses will be replaced after a day of wear. Objectives Primary Objective(s) The primary objective of this study are an evaluation of the clinical performance of logMAR visual acuity and subjective visual response. Study Endpoints Primary endpoints: logMAR visual acuity, and subjective visual response. Study Design The study is a bilateral, single masked, single-arm, 3-visit dispensing study. There will be one study treatment, with the subject being in the treatment for approximately 12-16 days. A total of approximately 36 eligible subjects will be targeted to complete the study (low Add hyperopes only). The subjects will be fit in the study lens and wear the optimized pair for 6-8 days. The primary endpoints of this study are logMAR visual acuity and subjective visual response. See the flow chart at the end of the synopsis table for the schematic of the study visits and procedures of main observations (Figure 1). Sample Size | Test Article(s) | |
| Schedules basis. Replacement Schedule: The lenses will be replaced after a day of wear. Objectives Primary Objective(s) The primary objective of this study are an evaluation of the clinical performance of logMAR visual acuity and subjective visual response. Study Endpoints Primary endpoints: logMAR visual acuity, and subjective visual response. Study Design The study is a bilateral, single masked, single-arm, 3-visit dispensing study. There will be one study treatment, with the subject being in the treatment for approximately 12-16 days. A total of approximately 36 eligible subjects will be targeted to complete the study (low Add hyperopes only). The subjects will be fit in the study lens and wear the optimized pair for 6-8 days. The primary endpoints of this study are logMAR visual acuity and subjective visual response. See the flow chart at the end of the synopsis table for the schematic of the study visits and procedures of main observations (Figure 1). Sample Size | Wear and Replacement | Wear Schedule: The lenses will be used on a daily disposable |
| Objectives Primary Objective(s) The primary objectives of this study are an evaluation of the clinical performance of logMAR visual acuity and subjective visual response. Primary endpoints: logMAR visual acuity, and subjective visual response. Study Design The study is a bilateral, single masked, single-arm, 3-visit dispensing study. There will be one study treatment, with the subject being in the treatment for approximately 12-16 days. A total of approximately 36 eligible subjects will be targeted to complete the study (low Add hyperopes only). The subjects will be fit in the study lens and wear the study lenses for 6-8 days then undergo optimization and wear the optimized pair for 6-8 days. The primary endpoints of this study are logMAR visual acuity and subjective visual response. See the flow chart at the end of the synopsis table for the schematic of the study visits and procedures of main observations (Figure 1). Sample Size A total of approximately 40 eligible subjects will be enrolled with 36 subjects targeted to complete. Study Duration The study will last approximately 2 months. Healthy male and female volunteers with presbyopia will be screened as per criteria outlined below. All volunteers will have baseline measurements taken to ensure eligibility. The baseline procedures will occur after inform consent has been obtained. For a detailed list of procedures see the time and events schedule listed below. Eligibility Criteria Potential subjects must satisfy all of the following criteria to be | _ | · · |
| Objectives Primary Objective(s) The primary objectives of this study are an evaluation of the clinical performance of logMAR visual acuity and subjective visual response. Primary endpoints: logMAR visual acuity, and subjective visual response. Study Design The study is a bilateral, single masked, single-arm, 3-visit dispensing study. There will be one study treatment, with the subject being in the treatment for approximately 12-16 days. A total of approximately 36 eligible subjects will be targeted to complete the study (low Add hyperopes only). The subjects will be fit in the study lens and wear the study lenses for 6-8 days then undergo optimization and wear the optimized pair for 6-8 days. The primary endpoints of this study are logMAR visual acuity and subjective visual response. See the flow chart at the end of the synopsis table for the schematic of the study visits and procedures of main observations (Figure 1). Sample Size A total of approximately 40 eligible subjects will be enrolled with 36 subjects targeted to complete. Study Duration The study will last approximately 2 months. Healthy male and female volunteers with presbyopia will be screened as per criteria outlined below. All volunteers will have baseline measurements taken to ensure eligibility. The baseline procedures will occur after inform consent has been obtained. For a detailed list of procedures see the time and events schedule listed below. Eligibility Criteria Potential subjects must satisfy all of the following criteria to be | | |
| The primary objectives of this study are an evaluation of the clinical performance of logMAR visual acuity and subjective visual response. Primary endpoints: logMAR visual acuity, and subjective visual response. Study Design The study is a bilateral, single masked, single-arm, 3-visit dispensing study. There will be one study treatment, with the subject being in the treatment for approximately 12-16 days. A total of approximately 36 eligible subjects will be targeted to complete the study (low Add hyperopes only). The subjects will be fit in the study lens and wear the study lenses for 6-8 days then undergo optimization and wear the optimized pair for 6-8 days. The primary endpoints of this study are logMAR visual acuity and subjective visual response. See the flow chart at the end of the synopsis table for the schematic of the study visits and procedures of main observations (Figure 1). Sample Size A total of approximately 40 eligible subjects will be enrolled with 36 subjects targeted to complete. Study Duration Anticipated Study Population The study will last approximately 2 months. Healthy male and female volunteers with presbyopia will be screened as per criteria outlined below. All volunteers will have baseline measurements taken to ensure eligibility. The baseline procedures will occur after inform consent has been obtained. For a detailed list of procedures see the time and events schedule listed below. Eligibility Criteria Potential subjects must satisfy all of the following criteria to be | Objectives | |
| clinical performance of logMAR visual acuity and subjective visual response. Primary endpoints: logMAR visual acuity, and subjective visual response. Study Design The study is a bilateral, single masked, single-arm, 3-visit dispensing study. There will be one study treatment, with the subject being in the treatment for approximately 12-16 days. A total of approximately 36 eligible subjects will be targeted to complete the study (low Add hyperopes only). The subjects will be fit in the study lens and wear the study lenses for 6-8 days then undergo optimization and wear the optimized pair for 6-8 days. The primary endpoints of this study are logMAR visual acuity and subjective visual response. See the flow chart at the end of the synopsis table for the schematic of the study visits and procedures of main observations (Figure 1). Sample Size Atoal of approximately 40 eligible subjects will be enrolled with 36 subjects targeted to complete. Study Duration Anticipated Study Population Healthy male and female volunteers with presbyopia will be screened as per criteria outlined below. All volunteers will have baseline measurements taken to ensure eligibility. The baseline procedures will occur after inform consent has been obtained. For a detailed list of procedures see the time and events schedule listed below. Eligibility Criteria Potential subjects must satisfy all of the following criteria to be | Objectives | |
| Study Design The study is a bilateral, single masked, single-arm, 3-visit dispensing study. There will be one study treatment, with the subject being in the treatment for approximately 12-16 days. A total of approximately 36 eligible subjects will be targeted to complete the study (low Add hyperopes only). The subjects will be fit in the study lens and wear the study lenses for 6-8 days then undergo optimization and wear the optimized pair for 6-8 days. The primary endpoints of this study are logMAR visual acuity and subjective visual response. See the flow chart at the end of the synopsis table for the schematic of the study visits and procedures of main observations (Figure 1). Sample Size A total of approximately 40 eligible subjects will be enrolled with 36 subjects targeted to complete. Study Duration The study will last approximately 2 months. Healthy male and female volunteers with presbyopia will be screened as per criteria outlined below. All volunteers will have baseline measurements taken to ensure eligibility. The baseline procedures will occur after inform consent has been obtained. For a detailed list of procedures see the time and events schedule listed below. Eligibility Criteria Potential subjects must satisfy all of the following criteria to be | | clinical performance of logMAR visual acuity and subjective |
| Study Design The study is a bilateral, single masked, single-arm, 3-visit dispensing study. There will be one study treatment, with the subject being in the treatment for approximately 12-16 days. A total of approximately 36 eligible subjects will be targeted to complete the study (low Add hyperopes only). The subjects will be fit in the study lens and wear the study lenses for 6-8 days then undergo optimization and wear the optimized pair for 6-8 days. The primary endpoints of this study are logMAR visual acuity and subjective visual response. See the flow chart at the end of the synopsis table for the schematic of the study visits and procedures of main observations (Figure 1). Sample Size A total of approximately 40 eligible subjects will be enrolled with 36 subjects targeted to complete. Study Duration The study will last approximately 2 months. Healthy male and female volunteers with presbyopia will be screened as per criteria outlined below. All volunteers will have baseline measurements taken to ensure eligibility. The baseline procedures will occur after inform consent has been obtained. For a detailed list of procedures see the time and events schedule listed below. Eligibility Criteria Potential subjects must satisfy all of the following criteria to be | | |
| The study is a bilateral, single masked, single-arm, 3-visit dispensing study. There will be one study treatment, with the subject being in the treatment for approximately 12-16 days. A total of approximately 36 eligible subjects will be targeted to complete the study (low Add hyperopes only). The subjects will be fit in the study lens and wear the study lenses for 6-8 days then undergo optimization and wear the optimized pair for 6-8 days. The primary endpoints of this study are logMAR visual acuity and subjective visual response. See the flow chart at the end of the synopsis table for the schematic of the study visits and procedures of main observations (Figure 1). Sample Size A total of approximately 40 eligible subjects will be enrolled with 36 subjects targeted to complete. Study Duration The study will last approximately 2 months. Anticipated Study Population Healthy male and female volunteers with presbyopia will be screened as per criteria outlined below. All volunteers will have baseline measurements taken to ensure eligibility. The baseline procedures will occur after inform consent has been obtained. For a detailed list of procedures see the time and events schedule listed below. Eligibility Criteria Potential subjects must satisfy all of the following criteria to be | Study Endpoints | Primary endpoints: logMAR visual acuity, and subjective visual |
| dispensing study. There will be one study treatment, with the subject being in the treatment for approximately 12-16 days. A total of approximately 36 eligible subjects will be targeted to complete the study (low Add hyperopes only). The subjects will be fit in the study lens and wear the study lenses for 6-8 days then undergo optimization and wear the optimized pair for 6-8 days. The primary endpoints of this study are logMAR visual acuity and subjective visual response. See the flow chart at the end of the synopsis table for the schematic of the study visits and procedures of main observations (Figure 1). Sample Size A total of approximately 40 eligible subjects will be enrolled with 36 subjects targeted to complete. Study Duration The study will last approximately 2 months. Anticipated Study Population Healthy male and female volunteers with presbyopia will be screened as per criteria outlined below. All volunteers will have baseline measurements taken to ensure eligibility. The baseline procedures will occur after inform consent has been obtained. For a detailed list of procedures see the time and events schedule listed below. Eligibility Criteria Potential subjects must satisfy all of the following criteria to be | | response. |
| schematic of the study visits and procedures of main observations (Figure 1). Sample Size A total of approximately 40 eligible subjects will be enrolled with 36 subjects targeted to complete. Study Duration The study will last approximately 2 months. Healthy male and female volunteers with presbyopia will be screened as per criteria outlined below. All volunteers will have baseline measurements taken to ensure eligibility. The baseline procedures will occur after inform consent has been obtained. For a detailed list of procedures see the time and events schedule listed below. Eligibility Criteria Potential subjects must satisfy all of the following criteria to be | Study Design | dispensing study. There will be one study treatment, with the subject being in the treatment for approximately 12-16 days. A total of approximately 36 eligible subjects will be targeted to complete the study (low Add hyperopes only). The subjects will be fit in the study lens and wear the study lenses for 6-8 days then undergo optimization and wear the optimized pair for 6-8 days. The primary endpoints of this study are logMAR visual |
| schematic of the study visits and procedures of main observations (Figure 1). Sample Size A total of approximately 40 eligible subjects will be enrolled with 36 subjects targeted to complete. Study Duration The study will last approximately 2 months. Healthy male and female volunteers with presbyopia will be screened as per criteria outlined below. All volunteers will have baseline measurements taken to ensure eligibility. The baseline procedures will occur after inform consent has been obtained. For a detailed list of procedures see the time and events schedule listed below. Eligibility Criteria Potential subjects must satisfy all of the following criteria to be | | See the flow chart at the end of the synonsis table for the |
| observations (Figure 1). A total of approximately 40 eligible subjects will be enrolled with 36 subjects targeted to complete. Study Duration The study will last approximately 2 months. Healthy male and female volunteers with presbyopia will be screened as per criteria outlined below. All volunteers will have baseline measurements taken to ensure eligibility. The baseline procedures will occur after inform consent has been obtained. For a detailed list of procedures see the time and events schedule listed below. Eligibility Criteria Potential subjects must satisfy all of the following criteria to be | | · |
| Sample Size A total of approximately 40 eligible subjects will be enrolled with 36 subjects targeted to complete. Study Duration The study will last approximately 2 months. Healthy male and female volunteers with presbyopia will be screened as per criteria outlined below. All volunteers will have baseline measurements taken to ensure eligibility. The baseline procedures will occur after inform consent has been obtained. For a detailed list of procedures see the time and events schedule listed below. Eligibility Criteria Potential subjects must satisfy all of the following criteria to be | | * = |
| with 36 subjects targeted to complete. Study Duration The study will last approximately 2 months. Healthy male and female volunteers with presbyopia will be screened as per criteria outlined below. All volunteers will have baseline measurements taken to ensure eligibility. The baseline procedures will occur after inform consent has been obtained. For a detailed list of procedures see the time and events schedule listed below. Eligibility Criteria Potential subjects must satisfy all of the following criteria to be | Sample Size | |
| Study Duration The study will last approximately 2 months. Healthy male and female volunteers with presbyopia will be screened as per criteria outlined below. All volunteers will have baseline measurements taken to ensure eligibility. The baseline procedures will occur after inform consent has been obtained. For a detailed list of procedures see the time and events schedule listed below. Eligibility Criteria Potential subjects must satisfy all of the following criteria to be | Sample Size | |
| Anticipated Study Population Healthy male and female volunteers with presbyopia will be screened as per criteria outlined below. All volunteers will have baseline measurements taken to ensure eligibility. The baseline procedures will occur after inform consent has been obtained. For a detailed list of procedures see the time and events schedule listed below. Eligibility Criteria Potential subjects must satisfy all of the following criteria to be | Study Duration | |
| Population screened as per criteria outlined below. All volunteers will have baseline measurements taken to ensure eligibility. The baseline procedures will occur after inform consent has been obtained. For a detailed list of procedures see the time and events schedule listed below. Eligibility Criteria Potential subjects must satisfy all of the following criteria to be | · | |
| baseline measurements taken to ensure eligibility. The baseline procedures will occur after inform consent has been obtained. For a detailed list of procedures see the time and events schedule listed below. Eligibility Criteria Potential subjects must satisfy all of the following criteria to be | 1 * | |
| procedures will occur after inform consent has been obtained. For a detailed list of procedures see the time and events schedule listed below. Eligibility Criteria Potential subjects must satisfy all of the following criteria to be | Горишноп | |
| For a detailed list of procedures see the time and events schedule listed below. Eligibility Criteria Potential subjects must satisfy all of the following criteria to be | | |
| listed below. Eligibility Criteria Potential subjects must satisfy all of the following criteria to be | | = - |
| Eligibility Criteria Potential subjects must satisfy all of the following criteria to be | | ± |
| | Fligibility Criteria | |
| | Lingionity Criteria | |

- 1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
- 2. The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
- 3. The subject must be at least 40 and not more than 70 years of age at the time of screening.
- 4. The subject's distance spherical component of their refraction must be in the range of +1.25 D to +3.75 D in each eye.
- 5. The subject's refractive cylinder must be -1.00 to -1.50 D in each eye.
- 6. The subject's ADD power must be in the range of +0.75 D to +1.50 D in each eye.
- 7. Subject's refractive cylinder axis must be within  $90^{\circ}\pm30^{\circ}$  or  $180^{\circ}\pm30^{\circ}$  in each eye.
- 8. The subject must have best corrected visual acuity of 20/20<sup>-3</sup> or better in each eye.
- 9. Subjects must own a wearable pair of spectacles if required for their distance vision.
- 10. The subject must already be wearing a presbyopic contact lens correction (e.g., reading spectacles over contact lenses, multifocal or monovision contact lenses, etc.) or if not respond positively to at least one symptom on the "Presbyopic Symptoms Questionnaire".

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

- 1. Currently pregnant or lactating.
- 2. Any active or ongoing ocular or systemic allergies that may interfere with contact lens wear.
- 3. Any active or ongoing systemic disease, autoimmune disease, or use of medication, which may interfere with contact lens wear. This may include, but not be limited to, diabetes, hyperthyroidism, Sjögren's syndrome, xerophthalmia, acne rosacea, Stevens-Johnson syndrome, and immunosuppressive diseases or any infectious diseases (e.g. hepatitis, tuberculosis).
- 4. Clinically significant (Grade 3 or 4) corneal edema, corneal vascularization, corneal staining, tarsal abnormalities or bulbar injection, or any other corneal or ocular abnormalities which would contraindicate contact lens wear.
- 5. Entropion, ectropion, extrusions, chalazia, recurrent styes, dry eye, glaucoma, history of recurrent corneal erosions.
- 6. Any previous, or planned, ocular or intraocular surgery (e.g.

| | radial keratotomy, PRK, LASIK, lid procedures, cataract surgery, retinal surgery, etc.). 7. A history of amblyopia, strabismus or binocular vision abnormality. 8. Any current ocular infection or inflammation. 9. Any current ocular abnormality that may interfere with contact lens wear. 10. Use of any of the following oral medications within 1 week prior to enrollment: oral retinoid isotretinoin (e.g. Accutane), oral tetracyclines, topical scopolamine, oral antihistamines (e.g., Chlor-Trimeton, and Benadryl), systemic steroids. 11. Use of any ocular medication, with the exception of rewetting drops. 12. History of herpetic keratitis. 13. Participation in any contact lens or lens care product clinical trial within 30 days prior to study enrollment. 14. Employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician). 15. Any known hypersensitivity or allergic reaction to Eye-Cept® |
|---|---|
| Disallowed | rewetting drop solution. Use of any prescription or over-the-counter (OTC) medications |
| Medications/Interventions | that may affect contact lens wear. |
| Measurements and<br>Procedures | logMAR Visual acuity and Subjective responses for vision using the CLUE questionnaire. |
| Microbiology or Other<br>Laboratory Testing | None |
| Study Termination | The occurrence of one or more Unanticipated Adverse Device Effect (UADE), or any SAE where relationship to study agent cannot be ruled out, may result in stopping further dispensing investigational product. In the event of a UADE or SAE, the Sponsor Medical Monitor may unmask the treatment regimen of subject(s) and may discuss this with the Principal Investigator before any further subjects are enrolled. |
| Ancillary Supplies/ Study-<br>Specific Materials | Eye-Cept® Rewetting drops and saline for storing worn lenses. |
| Principal Investigator(s) and Study Institution(s)/Site(s) | A full list of Principal Investigators, clinical sites, and institutions is kept separately from the Study Protocol and is included in the study Trial Master File. |

Figure 1: Study Flowchart



#### COMMONLY USED ABBREVIATIONS AND DEFINITIONS OF TERMS

ADD Plus Power Required For Near Use

ADE Adverse Device Effect

AE Adverse Event/Adverse Experience
BCVA Best Corrected Visual Acuity

BSCVA Best Spectacle Corrected Visual Acuity

CFR Code of Federal Regulations
CLUE Contact Lens User Experience

COAS Complete Ophthalmic Analysis System

COM Clinical Operations Manager CRA Clinical Research Associate

CRF Case Report Form

CRO Contract Research Organization

CT Center Thickness

D Diopter

DMC Data Monitoring Committee eCRF Electronic Case Report Form EDC Electronic Data Capture

ETDRS Early Treatment Diabetic Retinopathy Study

FDA Food and Drug Administration

GCP Good Clinical Practice

HIPAA Health Insurance Portability and Accountability Act

HIV Human Immunodeficiency Virus

IB Investigator's Brochure ICF Informed Consent Form

ICH International Council on Harmonization IDE Investigational Device Exemption IEC Independent Ethics Committee IRB Institutional Review Board

ISO International Organization for Standardization

ITT Intent-to-Treat

JJVC Johnson & Johnson Vision Care, Inc.

LC Limbus Center

LogMAR Logarithm of Minimal Angle of Resolution MedDRA<sup>©</sup> Medical Dictionary for Regulatory Activities

MOP Manual of Procedures

NIH National Institutes of Health

OD Right Eye

OHRP Office for Human Research Protections
OHSR Office for Human Subjects Research

OS Left Eye
OU Both Eyes

PD Protocol Deviation

PHI Protected Health Information

PI Principal Investigator

PIG Patient Instruction Guide PQC Product Quality Complaint PRO Patient Reported Outcome

QA Quality Assurance QC Quality Control

SAE Serious Adverse Event/Serious Adverse Experience

SAP Statistical Analysis Plan SAS Statistical Analysis System

SD Standard Deviation

SOP Standard Operating Procedure

UADE Unanticipated Adverse Device Effect

USADE Unanticipated Serious Adverse Device Effect

VA Visual Acuity

#### 1. INTRODUCTION AND BACKGROUND

Johnson & Johnson Vision recently launched a multifocal contact lens, 1-DAY ACUVUE Moist Multifocal. The lens is recommended for presbyopes who have -0.75 D of refractive cylinder. There is a considerable population of presbyopic patients who have greater than -0.75 D of cylinder, in one or both eyes. Currently there are a limited number of soft toric multifocal lenses available and they have limited success as evidenced by the very small market share. To meet this unmet need Johnson & Johnson Vision has undertaken a toric multifocal development program leveraging the Moist Multifocal optical design and adding toric correction and lens stabilization that is currently utilized in the 1-Day Moist for Astigmatism lens.

A previous study evaluating this novel multifocal toric lens was completed on hyperopic subjects and the lens displayed acceptable clinical performance. The population in that study was skewed toward the higher ADD subjects. The purpose of this study was to evaluate the same design in a low ADD hyperopic population.

#### 1.1. Name and Descriptions of Investigational Products

Investigational Product: Toric Multifocal Contact manufactured in etafilcon A material. Refer to Table 1 in Section 6.1 of the protocol.

#### 1.2. Intended Use of Investigational Products

The lenses are intended to correct refractive astigmatism, hyperopia and presbyopia. The lenses will be used in a population of presbyopes who have -1.00 D to -1.50 D of cylinder and add powers of +0.75 D to +1.50 D.

#### 1.3. Summary of Findings from Nonclinical Studies

All previous pre-clinical findings were deemed satisfactory prior to proceeding with clinical trials on humans. For the most comprehensive nonclinical information regarding JJVC Toric Multifocal Contact Lens manufactured in etafilcon A material refer to the latest version of the CR-6278 Investigator's Brochure.

#### 1.4. Summary of Known Risks and Benefits to Human Subjects

For the most comprehensive risk and benefit information regarding JJVC Toric Multifocal Contact Lens manufactured in etafilcon A material refer to the latest version of the CR-6278 Investigator's Brochure and Informed Consent.

## 1.5. Relevant Literature References and Prior Clinical Data Relevant to Proposed Clinical Study

| The toric multifocal contact lens system has been evaluated in clinical tria | als in |
|---|---|
| See summary details of the studies by | below. |
| In 57 subjects completed the study as cohort. The study was a Sing | _ |
| hyperopic presbyopes with against the rule astigmatism. Lenses were dispense | ed and worn for |
| approximately two weeks of wear. The mean binocular high luminance, high | contrast distance |
| acuity was -0.049 logMAR and near was 0.059 logMAR. There was one no | n-ocular adverse |
| event (sprained left toe) that was not related to the study lens. The subject comple | eted the study. |

In 19 subjects completed the study as cohort. The study was a Single-Arm study in hyperopic presbyopes who had with the rule astigmatism. Lenses were dispensed and worn for approximately two weeks of wear. The mean binocular high luminance, high contrast distance acuity was 0.066 logMAR and near was 0.103 logMAR. There was one serious adverse event that was reported that was non-ocular and not related to the study lens. The subject had cholecystitis and the event resolved 2 days after the event start date and the subject was permanently discontinued from the study.

In myopic presbyopes who had with or against the rule astigmatism. Lenses were dispensed and worn for approximately two weeks of wear. The mean binocular high luminance, high contrast distance acuity was -0.090 logMAR and near was 0.031 logMAR. There were two non-ocular adverse events, one serious adverse event that was reported that was non-ocular adverse events (upper respiratory tract infection and cold/allergy symptoms) that were not related to the study lenses. Both subjects completed the study.

In myopic presbyopes with astigmatism. Lenses were dispensed and worn for approximately two weeks of wear. The mean binocular high luminance, high contrast distance acuity was -0.101 logMAR and near was 0.024 logMAR. Two ocular events were reported by 1 subject during the study. The subject experienced non-significant irritation and redness of mild severity in both the eyes. Though the event resolved on the same day of occurrence without any treatment, the study lens was permanently discontinued and subject did not complete the study. The event was considered to be very likely related to the study treatment.

In the study in hyperopic presbyopes with astigmatism. Lenses were dispensed and worn for approximately two weeks of wear. The mean binocular high luminance, high contrast distance acuity was -0.023 logMAR and near was 0.103 logMAR. There was one non-ocular adverse event (nausea) that was determined to be not related to the study lenses.

#### 2. STUDY OBJECTIVES, ENDPOINTS AND HYPOTHESES

#### 2.1. Objectives

Primary Objective

The primary objectives of this study are an evaluation of the clinical performance of logMAR visual acuity and subjective visual response.

Secondary Objective Not applicable.

#### 2.2. Endpoints

Primary Endpoint

The primary endpoints of this study are logMAR visual acuity and subjective visual response.

Secondary Endpoint Not applicable.

Other Exploratory Endpoint(s) Not Applicable

## 2.3. Hypotheses

The following hypotheses will be tested throughout this investigation.

#### Primary Hypotheses

- 1. After 12-16 days of wear, the binocular bright, high contrast distance (4M) logMAR visual acuity of the test lens will be statistically better than +0.1 logMAR. This will be determined using ETDRS LogMAR acuity testing charts.
- 2. After 12-16 days of wear, the binocular bright, high contrast near (40cm) logMAR visual acuity of the test lens will be statistically better than +0.17 logMAR. This will be determined using Guillon/Poling LogMAR acuity testing charts.
- 3. After 12-16 days of wear, the PRO CLUE vision score for the test lenses will be statistically better than 32 points. This will be recorded by the subject using the CLUE follow-up questionnaire.

Secondary Hypotheses Not applicable.

Other Hypotheses Not applicable.

#### 3. TARGETED STUDY POPULATION

#### 3.1. General Characteristics

The population to be studied will consist of adapted contact lens wearers who have astigmatism in both eyes. Approximately 40 eligible subjects will be enrolled with 36 targeted to complete the study. Subjects will be targeted to be enrolled who have -1.00D to -1.50D of astigmatism in both eyes.

#### 3.2. Inclusion Criteria

Potential subjects must satisfy all of the following criteria to be enrolled in the study:

- 1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
- 2. The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
- 3. The subject must be at least 40 and not more than 70 years of age at the time of screening.
- 4. The subject's distance spherical component of their refraction must be in the range of +1.25 D to +3.75 D in each eye.
- 5. The subject's refractive cylinder must be -1.00 to -1.50 D in each eye.
- 6. The subject's ADD power must be in the range of +0.75 D to +1.50 D in each eye.
- 7. Subject's refractive cylinder axis must be within 90°±30° or 180°±30° in each eye.
- 8. The subject must have best corrected visual acuity of 20/20<sup>-3</sup> or better in each eye.
- 9. Subjects must own a wearable pair of spectacles if required for their distance vision.
- 10. The subject must already be wearing a presbyopic contact lens correction (e.g., reading spectacles over contact lenses, multifocal or monovision contact lenses, etc.) or if not respond positively to at least one symptom on the "Presbyopic Symptoms Questionnaire".

#### 3.3. Exclusion Criteria

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

- 1. Currently pregnant or lactating.
- 2. Any active or ongoing ocular or systemic allergies that may interfere with contact lens wear.
- 3. Any active or ongoing systemic disease, autoimmune disease, or use of medication, which may interfere with contact lens wear. This may include, but not be limited to, diabetes, hyperthyroidism, Sjögren's syndrome, xerophthalmia, acne rosacea, Stevens-Johnson syndrome, and immunosuppressive diseases or any infectious diseases (e.g. hepatitis, tuberculosis).
- 4. Clinically significant (Grade 3 or 4) corneal edema, corneal vascularization, corneal staining, tarsal abnormalities or bulbar injection, or any other corneal or ocular abnormalities which would contraindicate contact lens wear.
- 5. Entropion, extrusions, chalazia, recurrent styes, dry eye, glaucoma, history of recurrent corneal erosions.
- 6. Any previous, or planned, ocular or intraocular surgery (e.g. radial keratotomy, PRK, LASIK, lid procedures, cataract surgery, retinal surgery, etc.).
- 7. A history of amblyopia, strabismus or binocular vision abnormality.
- 8. Any current ocular infection or inflammation.
- 9. Any current ocular abnormality that may interfere with contact lens wear.
- 10. Use of any of the following oral medications within 1 week prior to enrollment: oral retinoid isotretinoin (e.g. Accutane), oral tetracyclines, topical scopolamine, oral antihistamines (e.g., Chlor-Trimeton, and Benadryl), systemic steroids.
- 11. Use of any ocular medication, with the exception of rewetting drops.
- 12. History of herpetic keratitis.

- 13. Participation in any contact lens or lens care product clinical trial within 30 days prior to study enrollment.
- 14. Employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician).
- 15. Any known hypersensitivity or allergic reaction to Eye-Cept® rewetting drop solution.

#### 3.4. Enrollment Strategy

Study subjects will be recruited from the Institution/clinical site's subject database and/or utilizing Independent Ethics Committee (IEC) or Institutional Review Board (IRB) approved materials.

#### 4. STUDY DESIGN AND RATIONALE

#### 4.1. Description of Study Design

The study is a bilateral, single masked, single-arm, 3-visit dispensing study. There will be one study treatment, with the subject being in the treatment for approximately 12-16 days. A total of approximately 36 eligible subjects will be targeted to complete the study (low Add hyperopes only). The subjects will be fit in the study lens and wear the study lenses for 6-8 days then undergo optimization and wear the optimized pair for 6-8 days. The primary end points are logMAR visual acuity and subjective visual response.

#### 4.2. Study Design Rationale

The study design is single-arm and the performance will be compared to previously set criteria for visual acuity and subjective vision response.

#### 4.3. Enrollment Target and Study Duration

A total of approximately 40 eligible subjects will be enrolled with 36 subjects targeted to complete. The study will last approximately 2 months.

#### 5. TEST ARTICLE ALLOCATION AND MASKING

#### **5.1.** Test Article Allocation

This study is a single-masked (subject masked), single-arm, dispensing clinical trial. Due to the nature of the study randomization is not required. All eligible subjects will be assigned to wear the same test article according to the lens wearing schedule.

#### 5.2. Masking

Masking will be used to reduce potential bias. Subjects will be unaware of the identity of the investigational product. Investigators and clinical site personnel involved in the data collection will not be masked as to the identity of the investigational product.

Under normal circumstances, the mask should not be broken until all subjects have completed the study and the database is finalized. Otherwise, the mask should be broken only if specific emergency treatment/course of action would be dictated by knowing the treatment status of the subject. In such cases, the Investigator may, in an emergency, contact the medical monitor. In the event the mask is broken, the Sponsor must be informed as soon as possible. The date, time, and reason for the unmasking must be documented in the subject record. The Investigator is also advised not to reveal the study treatment assignment to the clinical site or Sponsor personnel.

Subjects who have had their treatment assignment unmasked are expected to return for all remaining scheduled evaluations. Subjects who are discontinued may be replaced.

#### 5.3. Procedures for Maintaining and Breaking the Masking

The test articles mask shall not be broken unless information concerning the lens type is necessary for the urgent medical treatment of a subject. The Sponsor must be notified before the mask is broken.

When dispensing test articles, the following steps should be followed to maintain randomization codes:

- 1. Investigator or designee (documented on the Delegation Log) will consult the lens fitting schedule/randomization scheme to obtain the test article assignment for that subject prior to dispensing
- 2. Investigator or designee will record the subject's number on the appropriate line of the randomization scheme
- 3. Investigator or designee will pull the appropriate test articles from the study supply. All test articles that are opened, whether dispensed (placed/fit on eye or dispensed outside the clinical site) or not, must be recorded on the Test Article Accountability Log in the "Dispensed" section.

## 6. STUDY INTERVENTION

## 6.1. Identity of Test Articles

The following contact lenses will be used in this study:

Table 1: Test Articles

| | Test Lens |
|--------------------------------------|--------------------------------|
| Name | Investigational Toric |
| | Multifocal Contact Lens |
| Manufacturer | Johnson & Johnson |
| | Vision |
| Lens Material | etafilcon A with PVP |
| Nominal Base Curve @ 22°C | 8.5 |
| Nominal Diameter @ 22°C | 14.5 |
| Nominal Distance Powers (D) | +1.00 D to +4.00 D in |
| 22 | 0.25D steps |
| Nominal Cylinder Powers (D) and | -1.00 D cylinder with |
| Axes | 70°, 90°, 110°, 20°, |
| | 160°, 180° axes |
| Nominal ADD Power (D) | Low, Mid, High |
| Water Content | 58% |
| Center Thickness | 0.09 mm (-3.00 D) |
| Oxygen Permeability (Dk) | 23.8 x 10 <sup>-11</sup> (edge |
| 1000000000 | corrected). |
| Wear Schedule in Current Study | Daily Wear |
| Replacement Frequency | Daily Disposable |
| Packaging Form (vial, blister, etc.) | Blister |





#### 6.2. Ancillary Supplies/Products

The following solutions will be used in this study:

Table 2: Ancillary Supplies

| | Solution |
|---------------------------|-----------------|
| Calution Nama/Description | Eye-Cept® |
| Solution Name/Description | Rewetting Drops |
| Manufacturer | Optics |
| Waliufacturei | Laboratory |
| Preservative | Non-Preserved |

#### 6.3. Administration of Test Articles

Test articles will be dispensed to subject meeting all eligibility requirements, including any dispensing requirements set forth in this clinical protocol. Subjects will be dispensed an adequate supply of test articles to complete the study. Lost or damaged test articles may be replaced at the discretion of the Investigator and/or the Sponsor.

#### 6.4. Packaging and Labeling

The test articles will be packaged in blisters, glass vial, etc. as the primary packaging. The test article will be over-labeled to mask the subject to the identity of the lens. The test articles will be in plastic bags as the secondary packaging form.

The sample study label is shown below:



#### 6.5. Storage Conditions

Test articles will be maintained at ambient temperatures at the clinical site. Test articles must be kept under secure conditions.

#### 6.6. Collection and Storage of Samples

When possible, any lens or test article associated with an Adverse Events and/or a Product Quality Complaint must be retained and stored in a glass vial with moderate solution pending directions from the sponsor for potential return to JJVC.

#### 6.7. Accountability of Test Articles

JJVC will provide the Investigator with sufficient quantities of study articles and supplies to complete the investigation. The Investigator is asked to retain all lens shipment documentation for the test article accountability records.

Test article must be kept in a locked storage cabinet, accessible only to those assigned by the Investigator for dispensing. The Investigator may delegate this activity to authorized study site personnel listed on the Site Delegation Log. All test articles must be accounted. This includes:

- What was dispensed for the subject for trial fitting, to wear out of the office, or issued for the subject to replace appropriately between visits
- 2. What was returned to the Investigator unused
- 3. The number and reason for unplanned replacements

The Investigator will collect all unused test articles from the subjects at the end of the subject's participation. Subject returned unused test articles must be separated from the clinical study inventory of un-dispensed test articles, and must be labeled with the subject number and date of return. Following final reconciliation of test articles by the monitor, the Investigator or monitor will return all unused test articles to JJV.

If there is a discrepancy between the shipment documents and the contents, contact the study monitor <u>immediately.</u>

## 7. STUDY EVALUATIONS

## 7.1. Time and Event Schedule

Table 3: Time and Events

| Visit Information | Visit 1 | Visit 2 | Visit 3 |
|-----------------------------|------------|---------------|--------------|
| | Screening, | Treatment 1 | Treatment 1 |
| | Baseline, | Follow-up | Follow-up, |
| | Treatment | 3500 | Treatment 2 |
| | 1 | | |
| Time Point | Day 1 | Day $7 \pm 1$ | Day 7 ± 1 |
| | (Day 0) | From Visit 1 | from Visit 2 |
| Estimated Visit Duration | 2.5 hours | 1.0 hours | 1.5 hours |
| Statement of Informed | | | |
| Consent | X | | |
| Demographics | X | | |
| Medical | | | |
| History/Concomitant | | | |
| Medications/Review | X | X | X |
| Current Habitual | 31 | | |
| Correction | X | 5 | |
| Habitual Contact Lens | 0- | | |
| Information (if applicable) | X | 5 | |
| Contact Lens History (if | | | |
| applicable) | X | 5: | |
| Habitual Lens Wear Time | 01 | | |
| (if applicable) | X | 5: | |
| Screening | 0: | | |
| Inclusion/Exclusion | | | |
| Criteria | X | | |
| Ocular Symptoms | X | X | X |
| Entrance Distance and | | | |
| near Visual Acuity | X | X | X |
| Lens Removal (if | | | |
| applicable) | X | X | X |
| Keratometry | X | | |
| Subjective Sphero- | | | |
| Cylindrical Refraction | X | | |
| Near Add Determination | X | | |
| Ocular Dominance | X | | |
| Add Refinement | X | | |
| Near Visual Acuity | X | | |
| Slit Lamp Biomicroscopy | X | X | X |
| Baseline Inclusion/ | X | | |

| Visit Information | Visit 1 | Visit 2 | Visit 3 |
|---------------------------|------------|------------------|---------------|
| | Screening, | Treatment 1 | Treatment 1 |
| | Baseline, | Follow-up | Follow-up, |
| | Treatment | 150.00 | Treatment 2 |
| | 1 | | |
| Time Point | Day 1 | Day 7 ± 1 | Day $7 \pm 1$ |
| | (Day 0) | From Visit 1 | from Visit 2 |
| Estimated Visit Duration | 2.5 hours | 1.0 hours | 1.5 hours |
| Exclusion | | | |
| Lens Selection | X | X (if optimized) | |
| Right Lens Insertion | X | X (if optimized) | |
| Right Lens 1 Minute and 3 | | | |
| Minute Rotation | X | X (if optimized) | |
| Left Lens Insertion | X | X (if optimized) | |
| Left Lens 1 Minute and 3 | | | |
| Minute Rotation | X | X (if optimized) | |
| Lens Settling | X | X (if optimized) | |
| Toric Fit Assessment | Х | X | X |
| Subjective Lens Fit | | | |
| Assessment | X | X | X |
| Visual Satisfaction | X | X (if optimized) | |
| Subjective Acceptance | | X | X |
| Study Lens Distance and | | | |
| Near Visual Acuity | X | X | X |
| Over Refraction and | | | |
| Visual Acuity | X | X | |
| Lens Power Modification | | | |
| (if applicable) | X | 145 | |
| Insertion and Removal | | | |
| Training | X | la . | |
| Determination of | | | |
| Successful I/R | X | | |
| Determination of Lens | | | |
| Optimization | | X | |
| Lens Optimization (if | | | |
| required) | | X | |
| Insertion of Study Lenses | Х | X | |
| Post Fit Questionnaires | X | X | |
| Exit Snellen Distance and | | | |
| Near Visual Acuity | X | X | |
| Dispensing Criteria | X | X | |
| Subject Instructions | X | X | |
| Instruction Guide | x | ja<br>Na | |
| Lens Dispensing | X | X | |
| Schedule Follow-Up | x | X | |
| | • | | |

| Visit Information | Visit 1 | Visit 2 | Visit 3 |
|---|---|---|---|
| , 1510 111101111111111111111111111111111 | Screening, | Treatment 1 | Treatment 1 |
| | Baseline, | Follow-up | Follow-up, |
| | Treatment | | Treatment 2 |
| | 1 | | |
| Time Point | Day 1 | Day 7 ± 1 | Day 7 ± 1 |
| A A COLLEGE AND | (Day 0) | From Visit 1 | from Visit 2 |
| Estimated Visit Duration | 2.5 hours | 1.0 hours | 1.5 hours |
| Compliance | | X | X |
| Study Lens Wear Time | | X | X |
| Follow-up PRO and | | | |
| CLDEQ-8 Questionnaire | | X | X |
| Binocular Over Refraction | io | | X |
| Distance, Intermediate, | | | |
| and Near ETDRS | | | |
| LogMAR Visual Acuity | | | X |
| Collection of Unworn | | | |
| Lenses (if applicable) | | X | X |
| Study Completion | | | X |

## 7.2. Detailed Study Procedures

## VISIT 1

Subjects may report to the initial visit wearing their habitual contact lenses or spectacles (if required)

| | Visit 1: Screening | |
|---|---|---|
| Step | Procedure | Details |
| 1.1 | Statement of Informed<br>Consent | Each subject must read, understand, and sign the Statement of Informed Consent before being enrolled into the study. The Principal Investigator or his/her designee conducting the informed consent discussion must also sign the consent form. Note: The subject must be provided a signed |
| 1.2 | Demographics | copy of this document. Record the subject's year of birth, age, gender, race and ethnicity. |
| 1.3 | Medical History and<br>Concomitant<br>Medications | Questions regarding the subjects' medical history and concomitant medications. |
| 1.4 | Current Habitual<br>Correction | Record the subject's current habitual correct (i.e. Spectacles or Contact lenses) |
| 1.5 | Habitual Lenses (if applicable) | Questions regarding the subject's habitual lens type and parameters. |
| 1.6 | Contact Lens History<br>(If applicable) | Record the subject's correction type (i.e. monovision, multifocal, sphere with readers, etc.). |
| 1.7 | Wear time and<br>Comfortable Wear<br>time with Habitual<br>lenses (If applicable) | Record the subjects wear time and comfortable wear time with their habitual contact lenses. |
| 1.8 | Eligibility after<br>Screening | All responses to Screening Inclusion Criteria questions must be answered "yes" and all responses to Exclusion Criteria must be answered "no" for the subject to be considered eligible. If subject is deemed to be ineligible after screening, proceed to Final Evaluation and complete Subject Disposition. Refraction and Biomicroscopy forms are not required. |

| | Visit 1: Baseline | |
|------|-------------------|---------|
| Step | Procedure | Details |

| | | Visit 1: Baseline |
|---|---|---|
| Step | Procedure | Details |
| 1.9 | Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire. |
| 1.10 | Entrance Distance and<br>Near Visual Acuity | Distance and near Snellen visual acuity will be measured for each eye with the subject's habitual correction in place (if required). |
| | | For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be recorded to the nearest letter OD, OS and OU. |
| 1.11 | Lens Removal (If applicable) | Have the subject remove their habitual lenses and store in an approved storage solution. |
| 1.12 | Keratometry | Keratometry will be performed OD and OS and<br>the steep and flat dioptric power and<br>corresponding meridians recorded. |
| 1.13 | Subjective Sphero-<br>cylindrical Refraction | An optimal, binocular balanced distance spherocylindrical refraction will be performed. Record the refraction and distance visual acuity to the nearest letter. Note: Best distance visual acuity with sphero- |
| | | cylindrical refraction must be at least 20/20 <sup>-3</sup> in each eye for the subject to be eligible in the study. |
| 1.14 | Near ADD<br>Determination | The near reading addition will be determined using the binocular crossed cylinder technique (BCC) at 40 cm followed by optimization in a trial frame in step 1.16 below. |
| 1.15 | Ocular Dominance | Determine the distance ocular dominance with the best distance correction in place using a +1.00-blur test. If the results are equivocal use the sighting dominance test to determine the dominant eye used for the study. |
| 1.16 | ADD Refinement | Place the BCC result in the trial frame and refine<br>the near prescription with trial lenses (or<br>flippers) under binocular conditions. |
| 1.17 | Near Visual Acuity | Using the ETDRS 2000 Series Chart 1 or 2 near card placed at 40 cm. Record the near visual acuity OD, OS and OU at 40 cm. |
| 1.18 | Slit Lamp<br>Biomicroscopy | FDA Slit Lamp Classification Scale will be used to grade the findings and determine eligibility. |
| | | For the conjunctival redness 0.5-<br>unit increments will be used in the grading.<br>Corneal Staining Assessment will |

| | Visit 1: Baseline | |
|---|---|---|
| Step | Procedure | Details |
| | | be graded in 1.0 increments. If any of these slit lamp findings are Grade 3 or higher, the subject will be discontinued. If discontinued a final examination must be completed. |
| | | If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops or saline may be instilled. |
| 1.19 | Eligibility after<br>Baseline | All responses to Inclusion Criteria questions must be answered "yes" and all responses to Exclusion Criteria questions must be answered "no" for the subject to be considered eligible. If subject is deemed to be ineligible after |
| | | baseline, proceed to Final Evaluation and complete all forms. |

| | Visit 1: Treatment 1 Lens Fitting | |
|---|---|---|
| Step | Procedure | Details |
| 1.20 | Lens Selection | Select the lens power and axis based on the refraction and fitting guide for each eye. Record the test lens parameters (power and lot number). |
| 1.21 | Right Lens Insertion | Subjects will insert the right lens themselves. If the lens is uncomfortable, inspect for damage and remove, reinsert or replace as necessary. Damaged lenses will be stored in labeled vial with sterile saline, and clearly differentiated from the other worn lenses that will be shipped back to the Sponsor. Complete the Quality Product Complaint form. |
| 1.22 | Timed Settled for<br>Right Lens | The investigator will start a stopwatch as soon as the right lens is inserted. Note: All lenses in this study have scribe marks at 6 o'clock and 12 o'clock positions and rotation measurements are made relative to a vertical reference line. Record base nasal or base temporal rotation to the nearest degree. At one (1) minute after insertion: Record: 1. The rotational position to the nearest |

| | | degree |
|---|---|---|
| | | At three (3) minutes after insertion: Record: |
| | | 1. The rotational position to the nearest |
| 1.23 | Left Lens Insertion | degree Subjects will insert the left lens themselves. If |
| 1.23 | Left Lefts Hisertion | the lens is uncomfortable, inspect for damage |
| | | and remove, reinsert or replace as necessary. |
| | | Damaged lenses will be stored in labeled vial |
| | | with sterile saline, and clearly differentiated |
| | | from the other worn lenses that will be shipped |
| | | back to the Sponsor. Complete the Quality Product Complaint form. |
| 1.24 | Timed Settled for Left | The investigator will start a stopwatch as |
| | Lens | soon as the left lens is inserted. |
| | | Note: All lenses in this study have scribe |
| | | marks at 6 o'clock and 12 o'clock positions and rotation measurements are made relative |
| | | to a vertical reference line. |
| | | Record base nasal or base temporal rotation to |
| | | the nearest degree. |
| | | At one (1) minute after insertion: Record: |
| | | 1. The rotational position to the nearest |
| | | degree |
| | | At three (3) minutes after insertion: Record: |
| | | 1. The rotational position to the nearest |
| | | degree |
| 1.25 | Lens Settling | Allow the study lenses to settle for a minimum |
| 1.26 | Toric Fit | of 15 minutes. After lens settling, record: |
| 1.20 | Evaluation | • The rotational position to the nearest |
| | | degree |
| | | Lens stability with blink |
| | | Lens stability with eye versions |
| | | Toric fit acceptable or unacceptable Toric |
| | | lens fit will be unacceptable if lenses rotated |
| | | more than 40 degrees, or lens stability is worse |
| | | than 5 degrees movement with blink. If toric |
| | | fit is unacceptable, remove, store, and label the |
| | | lenses, and proceed to final evaluation. |
| 1.27 | Subjective Lens Fit | Evaluate and grade lens centration, primary gaze |

| | Assessment | movement, upgaze movement and tightness (push-up test). |
|---|---|---|
| | | <ul> <li>The subject should not proceed to wear the lenses if any of the following is observed:</li> <li>presence of limbal exposure (appearance of clear cornea) in any gaze</li> </ul> |
| | | <ul> <li>presence of edge lift</li> <li>presence of unacceptable movement<br/>(excessive or insufficient) in <u>all three</u><br/>movement categories (primary gaze, upgaze,<br/>and push-up).</li> </ul> |
| | | If either lens is deemed unacceptable, the subject will be discontinued from the study. Remove the lenses, perform a slit-lamp evaluation, and complete the Final Evaluation form. |
| 1.28 | Determine Visual<br>Satisfaction | Determine if the subject's vision is acceptable with the lenses. Allow the subject to look down a hallway or out of a window for distance vision assessments, and for them to read a book, magazine or similar for near vision. |
| 1.29 | Study Lens Distance<br>and Near Visual<br>Acuity | Measure the distance and near visual acuity OD, OS and OU to the nearest letter. Record the results. |
| | | <b>Note:</b> Use the ETDRS 2000 Series Chart 1 or 2 near card placed at 40 cm to measure the Near visual acuity. |
| 1.30 | Distance Over-<br>Refraction and<br>Distance Visual<br>Acuity | Perform a distance over-refraction OD and OS using loose lenses outside of the phoropter under ambient room illumination. The distance over-refraction may also be refined under binocular conditions. Record the results. The results of the distance over-refraction may also be checked for the impact on near vision under monocular and/or |
| 1.31 | Lens Power | binocular conditions. If the subject reports unsatisfactory vision, |
| | Modification (if applicable) | or is unable to obtain 20/30 distance visual acuity OU with the lenses than a modification must be attempted. If the subject reports satisfactory vision with the lenses a modification is not required however may at the Investigators discretion based upon their findings on the measured visual acuity and/or over- refraction. |

| _ | 1 | | , |
|---|---|---|---|
| | | Select the reason(s) for lens change (select all that apply): • The settled lens rotation is such that one of the other available lens cylinder axis would be better (use LARS rule to determine the replacement lens cylinder axis) • Power Modification needed • Unsatisfactory Vision • Other (specify reason) If one or both lenses are modified, repeat steps | |
| | | 1.20 through 1.30 for one or both eyes as | |
| | | appropriate. | |
| | | A maximum of <i>two</i> lens modifications are | |
| | | allowed. | |
| 1.32 | Post-Fit Questionnaire | The subject will evaluate the vision | |
| | | characteristics, comfort characteristics, handling | |
| | | characteristics, and visual symptoms of the study | |
| 1.33 | Insertion and | lenses using the PRO questionnaire. Neophytes and / or lapsed wearers who the | |
| 1.55 | Removal Training | investigator determines I/R training is required | |
| | (I/R) (if applicable) | will receive training on lens insertion, lens | |
| | (I/K) (II applicable) | removal, lens care and general contact lens | |
| | | safety information. | |
| | | Additional lenses may be used if necessary to | |
| | | complete the I&R training. Record the lens information on the Lens log and in EDC. | |
| | | information on the Bens log and in EBC. | |
| | | Note: Instruct the Neophytes / Lapsed wearer | |
| | | subjects to follow this wear schedule for the | |
| | | study lenses: | |
| | | Dispensing day: 6 hours of wear Day 1: 6-8 hours of wear | |
| | | Day 2: 6-10 hours of wear | |
| | | Day 3: 6-12 hours of wear | |
| | | Day 4 and subsequent days: 6 to all waking | |
| 1.21 | D | hours of wear | |
| 1.34 | Determination of I/R | The subject must be able to successfully insert and remove the contact lenses to be dispensed | |
| | Success (if | lenses and continue in the study. | |
| | applicable) | | |
| | | Note: If the subject is not able to successfully | |
| | | insert and remove the contact lenses the subject | |
| | | will be discontinued. | |
| | | Remove the lenses and complete the Final Evaluation. | |
| | | L variation. | |

| 1.35 | Exit Distance and | Distance and near Snellen visual acuity will |
|---|---|---|
| 1.55 | Near Visual Acuity | be measured for each eye to the nearest letter |
| | 1 (our visual riedity | with the study contact lenses in place. |
| | | For near measures use the ETDRS 2000 Series |
| | | Chart 1 or 2. The acuity will be recorded to the |
| | | nearest letter OD, OS and OU. |
| | | Note: The distance visual acuity must be at |
| 1.36 | Diananaina | least 20/30 OU for the lenses to be dispensed. The lenses will be dispensed for 6-8 days. |
| 1.30 | Dispensing | |
| | Criteria | Distance Snellen acuity equal to or better |
| | | than 20/30 OU |
| | | Subject must indicate that the vision is |
| | | acceptable. |
| | | Subject must indicate that the |
| | | comfort of the lenses is acceptable. |
| | | Lenses must have an acceptable toric and |
| | | general lens fit. |
| 1.37 | Subject Instructions | Instruct the Subject the following: |
| | | The lenses will be worn on a daily wear |
| | | basis. |
| | | Only enough lenses will be dispensed to the |
| | | subject to wear for the required number of |
| | | days until their follow-up visit. No additional |
| | | lenses will be dispensed. |
| | | A new lens will be opened and worn each |
| | | day. |
| | | Instruct the subject to bring back all unworn |
| | | study lenses. |
| | | No cleaning or disinfecting solutions will be |
| | | used. If determined necessary by the |
| | | Investigator sterile non-preserved rewetting |
| | | drops may be dispensed to be used as needed |
| | | for dryness. |
| | | Subjects will be instructed to wear lenses for |
| | | a minimum of 6 hours a day, every day |
| | | during the study. |
| | | Subjects will be instructed to wear their |
| | | glasses when not wearing the study lenses. |
| | | A patient instruction booklet will be |
| | | provided. |

| | | Note: In the event a lens is lost or damaged, the subject will return to the investigator site for replacement. As much as reasonably possible, a damaged lens should be returned to the investigational site and then returned to the Sponsor. If lens damage is present, complete the Product Quality Complaint Form. The lens will be stored in labeled vial with sterile saline, and returned to the Sponsor. |
|---|---|---|
| 1.38 | Schedule<br>Follow-up | The subject will be scheduled to return for their follow-up appointment in 7±1 day. |
| | | Note: To count the follow-up visit as a day of wear the Subject must have worn the study lenses for 6 hours prior to the visit. |

## VISIT 2

The subjects must present to Visit 2 wearing the study lenses. To be counted as a day of wear the lenses need to have been worn for at least six (6) hours prior to the visit.

| | Visit 2: Treatment 1 Follow-Up 1 | | |
|---|---|---|---|
| Step | Procedure | Details | |
| 2.1. | Adverse Events and<br>Concomitant<br>Medications Review | Review any changes to the subject's medical history or concomitant medications from the previous study visit. Record any changes, and any adverse events. | |
| 2.2. | Wear time and<br>Comfortable Wear<br>time (Study Lenses) | Record the average wearing time and comfortable wearing time with the study lenses. | |
| 2.3. | Compliance | Confirm compliance with the prescribed wear schedule. | |
| 2.4. | PRO and CLDEQ-8<br>Questionnaires | The subject will respond to the Follow-Up PRO and Dry Eye Questionnaires. | 200 |
| 2.5. | Subject Reported<br>Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire. | |
| 2.6. | Subjective Acceptance | Record whether the subjects distance and near vision with the lenses is acceptable. | |
| 2.7. | Entrance Distance and<br>Near Visual Acuity | Record the distance Snellen visual acuity with the contact lenses (OD, OS, and OU) to the nearest letter. For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be recorded to the nearest letter OD, OS and OU. | |
| 2.8. | Distance Over-<br>Refraction and<br>Distance Visual<br>Acuity | Perform a distance over-refraction OD and OS using loose lenses outside of the phoropter under ambient room illumination. The distance over-refraction may also be refined under binocular conditions. Record the results. The results of the distance over-refraction may also be checked for the impact on near vision under monocular and/or binocular conditions. | |
| 2.9. | Toric Fit<br>Evaluation | <ul> <li>After lens settling, record:</li> <li>The rotational position to the nearest degree</li> <li>Lens stability with blink</li> <li>Lens stability with eye versions</li> <li>Toric fit acceptable or unacceptable Toric lens fit will be unacceptable if lenses rotated more than 40 degrees, or lens stability is worse</li> </ul> | |

| Visit 2: Treatment 1 Follow-Up 1 | | | | | |
|---|---|---|--|--|--|
| Step | Procedure | Details | | | |
| | | than 5 degrees movement with blink. If toric | | | |
| | | fit is unacceptable, remove, store, and label the | | | |
| | | lenses, and proceed to final evaluation. | | | |
| 2.10. | Subjective Lens Fit | Evaluate and grade lens centration, primary gaze | | | |
| | Assessment | movement, upgaze movement and tightness | | | |
| | | (push-up test). | | | |
| | | The subject should not proceed to wear the | | | |
| | | lenses if any of the following is observed: | | | |
| | | SHARE | | | |
| | | <ul> <li>presence of limbal exposure (appearance of<br/>clear cornea) in any gaze</li> </ul> | | | |
| | | presence of edge lift | | | |
| | | presence of unacceptable movement | | | |
| | | (excessive or insufficient) in all three | | | |
| | | movement categories (primary gaze, upgaze, | | | |
| | | and push-up). | | | |
| | | If oither lang is decread an accountable the subject | | | |
| | | If either lens is deemed unacceptable, the subject will be discontinued from the study. Remove the | | | |
| | | lenses, perform a slit-lamp evaluation, and | | | |
| | | complete the Final Evaluation form. | | | |
| 2.11. | Determination of Lens | If the subjects vision is unacceptable for at | | | |
| | Optimization | least one distance or the Investigator determines | | | |
| | | that the visual acuity or over- refraction are not | | | |
| | | acceptable then a lens modification must be made. | | | |
| | | made. | | | |
| | | Up to <i>two</i> attempts at changes are permitted if | | | |
| | | necessary, in order to achieve an acceptable | | | |
| | | distance and near binocular performance for the | | | |
| | | subject. | | | |
| | | Follow the fitting guide allowing for at least | | | |
| | | 15 minutes of settling time between lens | | | |
| | | changes. | | | |
| 2.12. | Lens Optimization (if | Select the reason(s) for lens change (select | | | |
| | required) | all that apply): | | | |
| | | The settled lens rotation is such that one of the | | | |
| | | other available lens cylinder axis would be | | | |
| | | better (use LARS rule to determine the | | | |
| | | replacement lens cylinder axis). • Power Modification needed | | | |
| | | Unsatisfactory Vision | | | |
| | L | Clisatistactory vision | | | |
| | | Visit 2: Treatment 1 Follow-Up 1 | ting. |
|---|---|---|---|
| Step | Procedure | Details | |
| | | Other (specify reason) | |
| 2.13. | Lens Selection | Select the lens power, based on the Fitting | |
| | | Guide for each eye needing optimization. Record | |
| | | the test lens parameters (power and lot number). | |
| 2.14. | Lens Insertion | Subjects will insert the lens themselves. If the | |
| | | lens is uncomfortable, inspect for damage and | |
| | | remove, reinsert or replace as necessary. | |
| | | Damaged lenses will be stored in labeled vial | |
| | | with sterile saline, and clearly differentiated from | |
| | | the other worn lenses that will be shipped back to | |
| | | the Sponsor. Complete the Quality Product | |
| 2.15 | Time 1 Ca44 - 1 Ca - T | Complaint form. | 68 |
| 2.15. | Timed Settled for Lens | The investigator will start a stopwatch as soon as the lens is inserted. | |
| | | soon as the lens is inserted. | |
| | | Note: All lenses in this study have scribe | |
| | | marks at 6 o'clock and 12 o'clock positions | |
| | | and rotation measurements are made relative | |
| | | to a vertical reference line. | |
| | | Record base nasal or base temporal rotation to | |
| | | the nearest degree. | |
| | | At one (1) minute after insertion: Record: | |
| | | 1. The rotational position to the nearest | |
| | | degree | |
| | | At three (3) minutes after insertion: Record: | |
| | | 1. The rotational position to the nearest | |
| | | degree | |
| 2.16. | Lens Settling | Allow the study lenses to settle for a minimum of | |
| | and the second control of the second control | 15 minutes. | |
| 2.17. | Toric Fit | After lens settling, record: | |
| | Evaluation | <ul> <li>The rotational position to the nearest</li> </ul> | |
| | | degree | |
| | | Lens stability with blink | |
| | | Lens stability with eye versions | |
| | | Toric fit acceptable or unacceptable Toric | |
| | | lens fit will be unacceptable if lenses rotated | |
| | | more than 40 degrees, or lens stability is worse | |
| | | than 5 degrees movement with blink. If toric | |
| | | fit is unacceptable, remove, store, and label the | |
| | | lenses, and proceed to final evaluation. | |

| | | Visit 2: Treatment 1 Follow-Up 1 | ton to |
|---|---|---|---|
| Step | Procedure | Details | |
| 2.18. | Subjective Lens Fit<br>Assessment | Evaluate and grade lens centration, primary gaze movement, upgaze movement and tightness (push-up test). | |
| | | <ul> <li>The subject should not proceed to wear the lenses if any of the following is observed:</li> <li>presence of limbal exposure (appearance of clear cornea) in any gaze</li> <li>presence of edge lift</li> <li>presence of unacceptable movement (excessive or insufficient) in all three movement categories (primary gaze, upgaze, and push-up).</li> </ul> | |
| | | If either lens is deemed unacceptable, the subject will be discontinued from the study. Remove the lenses, perform a slit-lamp evaluation, and complete the Final Evaluation form. | |
| 2.19. | Determine Visual<br>Satisfaction | Determine if the subject's vision is acceptable with the lenses. Allow the subject to look down a hallway or out of a window for distance vision assessments, and for them to read a book, magazine or similar for near vision. | |
| 2.20. | Study Lens Distance<br>and Near Visual<br>Acuity | Measure the distance and near visual acuity (OD, OS and OU) to the nearest letter. Record the results. | |
| | | Note: Use the ETDRS 2000 Series Chart 1 or 2 near card placed at 40 cm to measure the Near visual acuity | |
| 2.21. | Distance Over-<br>Refraction and<br>Distance Visual<br>Acuity | Perform a distance over-refraction OD and OS using loose lenses outside of the phoropter under ambient room illumination. The distance over-refraction may also be refined under binocular conditions. Record the results. The results of the distance over-refraction may also be checked for the impact on near vision under monocular and/or binocular conditions. | |
| 2.22. | Additional Lens Power<br>Optimization (if<br>required) | If the subject reports unsatisfactory vision, or is unable to obtain 20/30 distance visual acuity OU with the lenses than a modification must be attempted. If the subject reports satisfactory vision with the lenses a modification is not | |

| | | Visit 2: Treatment 1 Follow-Up 1 |
|---|---|---|
| Step | Procedure | Details |
| | | required however may at the Investigators discretion based upon their findings on the measured visual acuity and/or over- refraction. |
| | | Select the reason(s) for lens change (select all that apply): • The settled lens rotation is such that one of the other available lens cylinder axis would be better (use LARS rule to determine the replacement lens cylinder axis) • Power Modification needed • Unsatisfactory Vision • Other (specify reason) |
| | | If one or both lenses are modified, repeat steps 2.13 through 2.21 for one or both eyes as appropriate. A maximum of <i>two</i> lens modifications are allowed. |
| 2.23. | Collection of unworn<br>lenses | Collect unworn lenses returned by the subject when lens power has been optimized. |
| | | If lens power was not changed allow the subject to use the unworn lenses dispensed at Visit 1 and dispense enough lenses of the same power to last the subject until their next visit. |
| 2.24. | Lens Removal | The optimized study lenses will be removed and discarded. |
| 2.25. | Slit Lamp<br>Biomicroscopy | FDA Slit Lamp Classification Scale will be used to grade the findings and determine eligibility. |
| | | For the conjunctival redness 0.5-unit increments will be used in the grading. Corneal Staining Assessment will be graded in 1.0 increments. If any of these slit lamp findings are Grade 3 or higher, the subject will be discontinued. If discontinued a final examination must be completed. |
| | | If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops or saline may be instilled. |
| 2.26. | Insertion of Study | Provide the subject with a new set of lenses |

| | Visit 2: Treatment 1 Follow-Up 1 | |
|---|---|---|
| Step | Procedure | Details |
| | Lenses | that match the power of the lenses that were |
| | | discarded in step 2.24 above. |
| 2.27. | Post-Fit Questionnaire | The subject will evaluate the vision |
| | | characteristics, comfort characteristics, handling |
| | | characteristics, and visual symptoms of the study |
| 2.28. | Exit Distance and | lenses using the PRO questionnaire. Distance and near Snellen visual acuity will |
| 2.28. | Near Visual Acuity | be measured OD, OS, and OU to the nearest |
| | Near Visual Activity | letter with the study contact lenses in place. |
| | | For near measures use the ETDRS 2000 Series |
| | | 2007 PA 1470 100 1 |
| | | Chart 1 or 2. The acuity will be recorded to the |
| | | nearest letter OD, OS and OU. |
| | | Note: The distance visual acuity must be at |
| 2.20 | D: | least 20/30 OU for the lenses to be dispensed. |
| 2.29. | Dispensing | The lenses will be dispensed for 6-8 days. |
| | Criteria | Distance Snellen acuity equal to or better<br>than 20/30 OU |
| | | Subject must indicate that the vision is |
| | | acceptable. |
| | | Subject must indicate that the |
| | | comfort of the lenses is acceptable. |
| | | Lenses must have an acceptable toric and |
| | | general lens fit. |
| 2.30. | Subject Instructions | Instruct the Subject the following: |
| | | The lenses will be worn on a daily wear |
| | | basis. |
| | | Only enough lenses will be dispensed to the |
| | | subject to wear for the required number of |
| | | days until their follow-up visit. No additional |
| | | lenses will be dispensed. |
| | | A new lens will be opened and worn each |
| | | day. |
| | | Instruct the subject to bring back all unworn |
| | | study lenses. |
| | | No cleaning or disinfecting solutions will be |
| | | used. If determined necessary by the |
| | | Investigator sterile non-preserved rewetting |
| | | drops may be dispensed to be used as needed |

| | Visit 2: Treatment 1 Follow-Up 1 | |
|---|---|---|
| Step | Procedure | Details |
| | | <ul> <li>Subjects will be instructed to wear lenses for a minimum of 6 hours a day, every day during the study.</li> <li>Subjects will be instructed to wear their glasses when not wearing the study lenses.</li> <li>Note: In the event a lens is lost or damaged, the subject will return to the investigator site for replacement. As much as reasonably possible, a damaged lens should be returned to the investigational site and then returned to the Sponsor. If lens damage is present, complete the Product Quality Complaint Form. The lens will be stored in labeled vial with sterile saline, and returned to the Sponsor.</li> </ul> |
| 2.31. | Schedule<br>Follow-up | The subject will be scheduled to return for their follow-up appointment in 7±1 day. Note: To count the follow-up visit as a day of wear the Subject must have worn the study lenses for 6 hours prior to the visit. |

# VISIT 3

The subjects must present to Visit 3 wearing the study lenses. To be counted as a day of wear the lenses need to have been worn for at least six (6) hours prior to the visit.

| | Visit 3: Treatment 1 Follow-Up 2 | | |
|---|---|---|---|
| Step | Procedure | Details | |
| 3.1. | Adverse Events and<br>Concomitant<br>Medications Review | Review any changes to the subject's medical history or concomitant medications from the previous study visit. Record any changes, and any adverse events. | |
| 3.2. | Wear time and<br>Comfortable Wear<br>time (Study Lenses) | Record the average wearing time and comfortable wearing time with the study lenses. | |
| 3.3. | Compliance | Confirm compliance with the prescribed wear schedule. | |
| 3.4. | PRO and CLDEQ-8<br>Questionnaires | The subject will respond to the Follow-Up PRO and Dry Eye Questionnaires. | 000 |
| 3.5. | Subject Reported<br>Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire. | |
| 3.6. | Subjective Acceptance | Record whether the subjects distance and near vision with the lenses is acceptable. | |
| 3.7. | Entrance Distance and<br>Near Visual Acuity | Record the distance Snellen visual acuity with the contact lenses (OD, OS, and OU) to the nearest letter. For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be recorded to the nearest letter OD, OS and OU. | |
| 3.8. | Binocular Distance<br>Over-refraction and<br>Distance Visual<br>Acuity | Perform a binocular over-refraction and record<br>the OD and OS results and distance visual acuity.<br>Note: No lens changes are allowed based on the<br>over-refraction. | |
| 3.9. | Toric Fit Evaluation | <ul> <li>After lens settling, record:</li> <li>The rotational position to the nearest degree</li> <li>Lens stability with blink</li> <li>Lens stability with eye versions</li> <li>Toric fit acceptable or unacceptable Toric lens fit will be unacceptable if lenses rotated more than 40 degrees, or lens stability is worse than 5 degrees movement with blink. If toric fit is unacceptable, remove, store, and label the lenses, and proceed to final evaluation.</li> </ul> | |
| 3.10. | Subjective Lens Fit | Evaluate and grade lens centration, primary gaze | |

| | | Visit 3: Treatment 1 Follow-Up 2 |
|---|---|---|
| Step | Procedure | Details |
| | Assessment | movement, upgaze movement and tightness (push-up test). |
| | | <ul> <li>The subject should not proceed to wear the lenses if any of the following is observed:</li> <li>presence of limbal exposure (appearance of clear cornea) in any gaze</li> <li>presence of edge lift</li> <li>presence of unacceptable movement (excessive or insufficient) in all three</li> </ul> |
| | | movement categories (primary gaze, upgaze, and push-up). If either lens is deemed unacceptable, the subject |
| | | will be discontinued from the study. Remove the lenses, perform a slit-lamp evaluation, and complete the Final Evaluation form. |
| 3.11. | Visual Performance<br>Distance (3M)<br>Intermediate (64 cm) | Visual performance will be recorded OD, OS, and OU for the following: Distance, Bright Illuminance |
| | Near (40 cm) | ETDRS Charts 3M-HC#1, HC#2, HC#3 and LC#1, LC#2 and LC#3 |
| | | Near, Bright Illuminance Reduced Guillon-Poling Charts High Contrast and Low Contrast Intermediate (64 cm) and Near (40 cm). |
| | | Distance, Dim Illuminance (with <u>Distance</u> goggles) |
| | | ETDRS Charts 3M-HC#4, HC#5, HC#6 Near, Dim Illuminance (with <u>Near</u> goggles) Reduced Guillon-Poling charts |
| | | High Contrast Intermediate (64 cm) and Near (40 cm). |
| | | Note: • The room illuminance must be between |
| | | 7.3 and 7.9 EV. • Distance, HC-1 Chart luminance Acceptable EV Range 10.5-10.7. |
| | | <ul> <li>Guillon-Poling, Near Chart Luminance<br/>Acceptable EV Range 10.8-11.1.</li> <li>Do not use the Mesopic filter for Dim</li> </ul> |

| 10.007-00- | 1 | Visit 3: Treatment 1 Follow-Up 2 |
|---|---|---|
| Step | Procedure | Details |
| a- a | | luminance (Dim luminance will be simulated by using the goggles). |
| 3.12. | Collection of unworn lenses (if applicable) | Collect unworn lenses returned by the subject. |
| 3.13. | Lens Removal | Have the subject remove the study lenses and store in saline in a labeled glass vial. Note: Lenses do not need to be stored in a refrigerator. |
| 3.14. | Slit Lamp<br>Biomicroscopy | FDA Slit Lamp Classification Scale will be used to grade the findings and determine eligibility. For the conjunctival redness 0.5-unit increments will be used in the grading. Corneal Staining Assessment will be graded in 1.0 increments. |
| | | If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops or saline may be instilled. |

#### FINAL EVALUATION

The final evaluation will ordinarily take place immediately following the last scheduled follow-up visit per the study protocol. It may also take place at any point the subject discontinues the study or is terminated from the study.

| | Final Evaluation | |
|---|---|---|
| Step | Procedure | Details |
| F.1 | Subjective<br>spherocylindrical<br>Refraction | An optimal, binocular balanced distance sphero-<br>cylindrical refraction will be performed. Record<br>the refraction and distance visual acuity to the<br>nearest letter. |
| F.2 | Final Exam Form | Indicate if the subject completed the study successfully. If subject discontinued from the study, indicate the reason. |

#### 7.3. Unscheduled Visits

If, during the investigation, a subject requires an unscheduled visit to the clinical site, the following information will be collected at a minimum:

- Chief complaint prompting the visit. If the reason is an adverse event, the applicable eCRF for the adverse event must be completed and subject record completed as appropriate
- Date and time of the visit and all procedures completed at the unscheduled visit
- Review of adverse event and concomitant medications
- Documentation of any test article dispensed or collected from the subject, if applicable
- Slit lamp findings (using the Slit Lamp Classification Scale)

If the Investigator withdraws a subject from the study, the final study visit case report forms must be completed indicating the reason(s) why the subject was withdrawn. The subject record must be completed documenting the date and primary reason for withdrawal and the study CRA notified.

Any ocular and non-ocular Adverse Events that are ongoing at the time of the study visit will be followed by the Investigator, within licensure, until they have resolved, returned to pre-treatment status, stabilized, or been satisfactorily explained. If further treatment i.e., beyond licensure is required, the subject will be referred to the appropriate health care provider.

The following information will be collected during an unscheduled visit.

| | Unscheduled Visit | |
|---|---|---|
| Step | Procedure | Details |
| U.1 | Chief Complaints | Record the subject's chief complaints for reasons for the unscheduled visit. |
| U.2 | Adverse Events and<br>Concomitant<br>Medications Review | Review any changes to the subject's medical history or concomitant medications from the previous study visit. Record any changes, and any adverse events. |

| | | Unscheduled Visit | |
|---|---|---|---|
| Step | Procedure | Details | |
| U.3 | Subject Reported | Subjects will respond to a verbal open-ended | # · |
| U.4 | Ocular Symptoms Entrance Visual | symptoms questionnaire. Record the entrance distance and near visual | _ |
| 0.4 | Acuity | acuity (OD, OS and OU) to the nearest letter. | |
| | Tieury | details (62), 65 and 66) to the nearest tetter. | |
| | | For near measures use the ETDRS 2000 Series | |
| | | Chart 1 or 2. The acuity will be recorded to the | |
| | | nearest letter OD, OS and OU. | _ |
| U.5 | Subjective Sphero- | An optimal, binocular balanced distance sphero- | |
| | cylindrical Refraction | cylindrical refraction will be performed. | |
| | | Record the refraction and distance visual acuity | |
| | | to the nearest letter. | |
| U.6 | Slit Lamp | FDA Slit Lamp Classification Scale will be used | |
| | Biomicroscopy | to grade the findings and determine eligibility. | |
| | | For the conjunctival redness 0.5- | |
| | | unit increments will be used in the grading. | |
| | | Corneal Staining Assessment will | |
| | | be graded in 1.0 increments. | |
| | | If the clearance of the fluorescein needs to be | |
| | | expedited, preservative-free rewetting drops or | |
| | | saline may be instilled. | |
| U.7 | Lens Dispensing | Additional study lenses may be dispensed when | |
| DATES - DATES DA | 2000 W 10 | required. | |
| U.8 | Toric Fit | After lens settling, record: | |
| | Evaluation | The rotational position to the nearest | |
| | | degree | |
| | | Lens stability with blink | |
| | | Lens stability with eye versions The formula in the stable in the | |
| | | Toric fit acceptable or unacceptable Toric | |
| | | lens fit will be unacceptable if lenses rotated | |
| | | more than 40 degrees, or lens stability is worse | |
| | | than 5 degrees movement with blink. If toric | |
| | | fit is unacceptable, remove, store, and label the | |
| *** | 19-14 P | lenses, and proceed to final evaluation. | |
| U.9 | Subjective Lens Fit | Evaluate and grade lens centration, primary gaze | |
| | Assessment | movement, upgaze movement and tightness (push-up test). | |
| | | (push up test). | |
| | | The subject should not proceed to wear the | |

| | Unscheduled Visit | |
|---|---|---|
| Step | Procedure | Details |
| | | lenses if any of the following is observed: • presence of limbal exposure (appearance of clear cornea) in any gaze • presence of edge lift • presence of unacceptable movement (excessive or insufficient) in all three movement categories (primary gaze, upgaze, and push-up). If either lens is deemed unacceptable, the subject will be discontinued from the study. Remove the lenses, perform a slit-lamp evaluation, and complete the Final Evaluation form. |
| U.10 | Exit Visual Acuity | Record the entrance distance and near visual acuity (OD, OS and OU) to the nearest letter. For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be recorded to the nearest letter OD, OS and OU. |

# 7.4. Laboratory Procedures

Not Applicable.

# 8. SUBJECTS COMPLETION/WITHDRAWAL

# 8.1. Completion Criteria

Subjects are considered to have completed the study if they:

- · provided informed consent
- they are eligible
- completed all visits

# 8.2. Withdrawal/Discontinuation from the Study

A subject will be withdrawn from the study for any of the following reasons:

- Subject death during the study period
- Subject withdrawal of consent
- Subject not compliant to protocol
- Subject lost to follow-up
- Subject no longer meets eligibility criteria (e.g. the subject becomes pregnant)
- Subject develops significant or serious adverse events causing discontinuation of study lens wear
- Subjects who have experienced a Corneal Infiltrative Event (CIE)

- Investigator's clinical judgment regarding the subject safety reasons (that it is in the best interest of the subject to stop treatment)
- Subject missed two consecutive study visits
- Subject not compliant with study lens wear schedule
- Subject not successfully dispensed due to lack of efficacy and safety including poor vision, poor comfort or unacceptable fit

For discontinued subjects, the Investigator will:

- Complete the current visit (scheduled or unscheduled)
- Complete the Final Evaluation, indicating the reason that the subject was discontinued from the study
- Record the spherocylindrical refraction with best corrected distance visual acuity
- Collect used test article(s) (worn or brought to the visit) from the subject and discard them, unless otherwise stated in Section 7.2
- Collect all unused test article(s) from the subject

An additional subject may be enrolled if a subject discontinues from the study prematurely.

In cases where a subject is lost to follow-up, every possible effort must be made to contact the subject and determine the reason for discontinuation/withdrawal. The measures taken to follow up must be documented including two written attempts and a certified letter (or equivalent) as the final attempt.

#### 9. PRE-STUDY AND CONCOMITANT INTERVENTION/MEDICATION

Concomitant medications will be documented during screening and updated during the study. Disallowed medications and therapies are medications or therapies that contraindicate contact lens wear. See the Exclusion criteria for specific details.

#### 10. DEVIATIONS FROM THE PROTOCOL

Investigator will notify study sponsor upon identification of a protocol deviation. Major protocol deviations must be reported to the sponsor within 24 hours after discovery of the protocol deviation. The Investigator will report deviations per IRB/IEC requirements. All deviations will be tracked and corrective actions implemented as appropriate.

If it becomes necessary for the Investigator to implement a deviation in order to eliminate an immediate hazard to the trial subject, the Investigator may implement the deviation immediately without notification to the sponsor. Within 24 hours after the implemented deviation, the Investigator must notify and provide the rationale to the Sponsor and, as required, the IEC/IRB.

## 11. STUDY TERMINATION

The occurrence of one or more Unanticipated Serious Adverse Device Effect (USADE), or any SAE where the relationship to study agent cannot be ruled out, may result in stopping further

dispensing of test article. In the event of a USADE or SAE, the Sponsor may unmask the treatment regimen for the subject(s) and will discuss this with the Investigator before any further subjects are enrolled.

The Sponsor will determine when a study will be stopped. The Principal Investigator always has the discretion to initiate stopping the study based on patient safety or if information indicates the study's results are compromised.

JJVC reserves the right to terminate the study at any time for any reason. Additionally, the IEC/IRB reserves the right to terminate the study if an unreasonable risk is determined. The study can be terminated by the Principal Investigator at the individual clinical site due to specific clinical observations, if in their opinion, after a discussion with JJVC, it is determined that it would be unwise to continue at the clinical site.

JJVC (and the IEC/IRB and DMC, if applicable) will evaluate all adverse events. If it is determined that an adverse event presents an unreasonable risk, the investigation, or that part of the investigation presenting the risk, will be terminated, as soon as possible.

Should the study be terminated (either prematurely or as scheduled), the Investigator will notify the IEC/IRB and Regulatory Authority as required by local regulatory requirements.

# 12. PROCEDURE FOR HANDLING PRODUCT QUALITY COMPLAINTS

A Product Quality Complaint (PQC) refers to any written, electronic, or oral communication that alleges deficiencies related to the identity, quality, durability, reliability, safety, effectiveness or performance of test articles after they have been released for clinical trial use.

Potential complaints may come from a variety of sources including but not limited to subjects, clinical research associates (CRA), clinical operations managers (COM), medical monitors, and site personnel, etc. The following are not considered product quality complaints:

- Subject satisfaction inquiries reported via "Subjective Questionnaires" and "Patient Reported Outcomes (PRO)"
- Clinical test articles that are stored improperly or damaged after receipt at the investigational site
- Lens replacements that occur due to drops/fall-outs
- Damage deemed by clinicians or clinical staff to be caused by handling by the user, and not indicative of a quality deficiency (i.e. tears, rips, etc.), only in situations where there is no deficiency alleged by the subject

Within 24 hours of site personnel becoming aware that a PQC has occurred, the PQC must be recorded in the EDC system, which will trigger an automatic email notification to the appropriate COM/CRA and Clinical QA representative. In cases where the EDC system in use is not configured to send automatic notifications or when an EDC system is not used, the COM/CRA is responsible for notifying Clinical QA upon discovery that a PQC has occurred.

Upon receipt of the EDC notification, the COM/CRA will contact the study site to collect additional information which will include:

- Date the complaint was received/recorded in the EDC System (Date of Sponsor Awareness)
- Who received the complaint
- Study number
- Clinical site information (contact name, site ID, telephone number)
- Lot number(s)
- Unique Subject Identifier(s)
- Indication of who first observed complaint (site personnel or subject)
- OD/OS indication, along with whether the lens was inserted
- Any related AE number if applicable
- Detailed complaint description (scheduled/unscheduled visit, wear time, symptoms, resolution of symptoms, etc.)
- Eye Care Provider objective (slit lamp) findings if applicable
- Confirmation of product availability for return (and tracking information, if available), or rationale if product is not available for return

Once a complaint is received, it will be assessed by the COM, CRA, or trained site personnel to determine if it is an Adverse Event/Serious Adverse Event (AE/SAE). If the complaint results in an AE/SAE, the COM/CRA, or trained site personnel will follow Section 13 of this protocol. If the AE/SAE was potentially the result of a product quality related deficiency, these procedures also applies and will be executed in parallel.

In some cases, a PQC form may be generated in EDC by the site in error. In this event, the PQC forms will be marked "Intentionally Left Blank" or "ILB". Justification for ILB must be documented.

#### 13. ADVERSE EVENTS

#### 13.1. Definitions and Classifications

**Adverse Event (AE)** – An AE is "any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the investigational medical device.

*Note 1* to entry: This definition includes events related to the investigational medical device or the comparator.

*Note 2* to entry: This definition includes events related to the procedures involved.

*Note 3* to entry: For users or other persons, this definition is restricted to events related to investigational medical devices."<sup>1</sup>

An AE includes any condition (including a pre-existing condition) that:

- 1. Was not present prior to the study, but appeared or reappeared following initiation of the study
- 2. Was present prior to the study, but worsened during the study. This would include any condition resulting from concomitant illnesses, reactions to concomitant medications, or progression of disease states
- 3. Pregnancy must be documented as an adverse event and must be reported to the clinical monitor and to the Sponsor immediately upon learning of the event

# **Serious Adverse Event (SAE)** – An SAE is any untoward medical occurrence that:

- Results in death
- Is life threatening
- Requires in-patient hospitalization or prolongation of existing hospitalization
- Results in persistent or significant disability/incapacity (e.g., a sight threatening event, a significant persistent or permanent change, impairment, damage, or disruption to the subject's body)
- Is a congenital anomaly/birth defect
- Requires intervention to prevent permanent damage (the use of the test article resulting in a condition which requires medical or surgical intervention to preclude permanent impairment of the body structure or a body function). Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered an SAE when, based upon appropriate medical judgment, they may jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the outcomes listed in the above definition

Diagnoses and conditions that are considered Ocular Serious Adverse Events include, but not limited to:

- Microbial Keratitis (MK)
- Iritis (including cells in the anterior chamber)
- Permanent decrease in best spectacle corrected visual acuity equivalent to 2 acuity lines or greater
- Central Corneal Opacity
- Central Corneal Neovascularization
- Uveitis
- Endophthalmitis
- Hypopyon
- Hyphemia
- Penetration of Bowman's Membrane
- Persistent Epithelial Defect
- Limbal cell Damage leading to Conjunctivalization

**Significant Adverse Events** – Those events that are usually symptomatic and warrant discontinuation (temporary or permanent) of the test article (excluding Serious Adverse Events).

Diagnoses and conditions that are considered Ocular Significant Adverse Events include, but not limited to the following:

- Contact Lens Induced Peripheral Ulcer (CLPU)
- Significant Infiltrative Events (SIE)
- Superior Epithelial Arcuate Lesions (SEALs)
- Any Temporary Loss of > 2 Lines of BSCVA
- Other grade 3 or higher corneal findings, such as abrasions or edema
- Non-contact lens related corneal events e.g. Epidemic Keratoconjunctivitis (EKC)
- Asymptomatic Corneal Scar
- Any corneal event which necessitates temporary lens discontinuation > 2 weeks

**Non-Significant Adverse Events** – Those conditions that are usually asymptomatic and usually do not warrant discontinuation (temporary or permanent) of the test article. However, the Investigator may choose to treat as a precautionary measure.

Diagnoses and conditions that are considered Ocular Non-Significant Adverse Events include, but not limited to the following:

- Non-significant Infiltrative Event (NSIE)
- Contact Lens Papillary Conjunctivitis (CLPC)
- Superficial Punctate Keratitis (SPK)
- Conjunctivitis: Bacterial, Viral, Allergic
- Blepharitis
- Meibomianitis
- Contact Dermatitis
- Localized Allergic Reactions
- Any corneal event not explicitly defined as serious or significant adverse event, which necessitates temporary lens discontinuation < 2 weeks

**Adverse Device Effect (ADE)** – An ADE is an "adverse event related to the use of an investigational medical device.

*Note 1* to entry: This definition includes adverse events resulting from insufficient or inadequate instructions for use, deployment, implantation, installation, or operation, or any malfunction of the investigational medical device.

*Note 2* to entry: This definition includes any event resulting from use error or from intentional misuse of the investigational medical device."<sup>1</sup>

Unanticipated Adverse Device Effect (UADE) – Any serious adverse effect on health or safety or any life-threatening problem or death caused by, or associated with, the test article, if that effect, problem, or death was not previously identified in nature, severity, or degree of incidence in the investigational plan, Investigator's Brochure or protocol, or any other unanticipated serious problem associated with the test article that relates to the rights, safety and welfare of subjects.

## 13.2. Assessing Adverse Events

In conjunction with the medical monitor, the Investigator will evaluate adverse events to ensure the events are categorized correctly. Elements of categorization will include:

- Seriousness/Classifications (see definition in Section 13.1)
- Causality or Relatedness i.e. the relationship between the test article, study treatment or study procedures and the adverse event (not related; unlikely related; possibly related; related see definition in Section 13.2.1)
- Adverse Event Severity Adverse event severity is used to assess the degree of intensity of the adverse event (mild; moderate; severe for all events see definition in Section 0)
- Outcome not recovered or not resolved; recovering or resolving; recovered or resolved with sequelae; recovered or resolved; death related to adverse event; unknown
- Actions Taken none; temporarily discontinued; permanently discontinued; other

# 13.2.1. Causality Assessment

Causality Assessment – A determination of the relationship between an adverse event and the test article. The test article relationship for each adverse event should be determined by the investigator using these explanations:

- Not Related- An adverse event that is not related to the use of the test article, study treatment or study procedures
- Unlikely Related An adverse event for which an alternative explanation is more likely, e.g. concomitant treatment, concomitant disease(s), or the relationship of time suggests that a causal relationship is not likely
- Possibly Related An adverse event that might be due to the use of the test article, or to the study treatment or study procedures. An alternative explanation, e.g. concomitant treatment, concomitant disease(s), is inconclusive. The relationship in time is reasonable. Therefore, the causal relationship cannot be excluded
- Related An adverse event that is listed as a possible adverse effect (device) or adverse reaction (drug) and cannot be reasonably explained by an alternative explanation, e.g. concomitant treatment of concomitant disease(s). The relationship in time is very suggestive, e.g. it is confirmed by de-challenge and re-challenge

#### 13.2.2. Severity Assessment

**Severity Assessment** – A qualitative assessment of the degree of intensity of an adverse event as determined by the Investigator or reported to him/her by the subject. The assessment of severity is made irrespective of test article, study treatment or study procedure relationship or seriousness of the event and should be evaluated according to the following scale:

- Mild Event is noticeable to the subject, but is easily tolerated and does not interfere with the subject's daily activities
- Moderate Event is bothersome, possible requiring additional therapy, and may interfere with the subject's daily activities
- Severe Event is intolerable, necessitates additional therapy or alteration of therapy and interferes with the subject's daily activities

## 13.3. Documentation and Follow-Up of Adverse Events

The recording and documenting of adverse events (ocular and non-ocular) begins when the subjects are exposed to the test article, study treatment or study procedure. Adverse events reported before the use of test article, start of study treatment, or study procedures will be recorded as medical history. However, if the condition deteriorates at any time during the study it will be recorded and reported as an AE. Untoward medical events reported after the subject's exit from the study will be recorded as adverse events at the discretion of the Investigator.

Upon finding an adverse event, the Principal Investigator will document the condition in the subject record and in the eCRFs. He/she will complete the Adverse Event /eCRF.

Complete descriptions of all adverse events must be available in the subject record. All Adverse Events including local and systemic reactions not meeting the criteria for "serious adverse events" shall be captured on the appropriate case report form or electronic data system. All adverse events occurring while the subject is enrolled in the study must be documented appropriately regardless of relationship.

It is the Investigator's responsibility to maintain documentation of each reported adverse event. All adverse events will be followed in accordance with applicable licensing requirements. Such documentation will include the following:

- Adverse event (diagnosis not symptom)
- Drawings or photographs (where appropriate) that detail the finding (e.g., size, location, and depth, etc.)
- Date the clinical site was notified
- Date and time of onset
- Date and time of resolution
- Adverse event classification, severity, and relationship to test articles, as applicable
- Treatment regimen instituted, including concomitant medications prescribed, in accordance with applicable licensing requirements
- Any referral to another health care provider if needed
- Outcome, ocular damage (if any)
- Likely etiology
- Best corrected visual acuity at the discovery of the event and upon conclusion of the event

In addition, if an infiltrate(s) is present, he/she will complete the Corneal Infiltrate Assessment eCRF. Where necessary, a culture of the corneal lesion will be collected to determine if the infection is microbial in nature. If cultures are collected, the date of culture collection and laboratory utilized will be recorded.

Changes in the severity of an AE shall be documented to allow an assessment of the duration of the event at each level of intensity to be performed. Adverse events characterized as intermittent require documentation of the onset and duration of each episode. Changes in the assessment of relationship to the Test Article shall also be clearly documented.

Subjects who present with an adverse event shall be followed by the Investigator, within licensure, until all signs and symptoms have returned to pre-treatment status, stabilized, or been satisfactorily resolved. If further treatment beyond licensure is required, the patient will be referred to the appropriate health care provider. The Investigator will use his/her clinical judgment as to whether a subject reporting with an adverse event will continue in the study. If a subject is discontinued from the study, it will be the responsibility of the Investigator to record the reason for discontinuation. The Investigator will also document the adverse event appropriately and complete the Adverse Event eCRF. Any subjects with ongoing adverse events related to the test article, study treatment or study procedures, as of the final study visit date, should be followed to resolution of the adverse event or until referral to an appropriate health care provider, as recommended by the Investigator. Non-ocular adverse events that are not related to the test article, study treatment, or study procedures may be recorded as "ongoing" without further follow-up.

# 13.4. Reporting Adverse Events

The Investigator will notify the Sponsor of an adverse event by e-mail, facsimile, or telephone as soon as possible and no later than 24 hours from discovery for any serious /significant adverse events, and 2 days from discovery for any non-significant adverse event. In addition, a written report will be submitted by the Principal Investigator to the IEC/IRB according to their requirements (Section 13.4.2). The report will comment whether the adverse event was considered to be related to the test article, study treatment or study procedures.

## 13.4.1. Reporting Adverse Events to Sponsor

#### **Serious/Significant Adverse Events**

The Investigator will inform the sponsor of all serious/significant adverse events occurring during the study period as soon as possible by e-mail, fax, or telephone, but no later than 24 hours following discovery of the event. The Investigator is obligated to pursue and obtain information requested by the Sponsor in addition to that information reported on the eCRF. All subjects experiencing a serious/significant adverse event must be followed up and all outcomes must be reported.

When medically necessary, the Investigator may break the randomization code to determine the identity of the treatment that the subject received. The Sponsor and study monitor should be notified prior to unmasking the test articles.

In the event of a serious/significant adverse event, the Investigator must:

- Notify the Sponsor immediately
- Obtain and maintain in the subject's records all pertinent medical information and medical judgment for colleagues who assisted in the treatment and follow-up of the subject
- Provide the Sponsor with a complete case history which includes a statement as to whether the event was or was not related to the use of the test article
- Notify the IEC/IRB as required by the IEC/IRB reporting procedure according to national regulations

# **Unanticipated (Serious) Adverse Device Effect (UADE)**

In the event of an Unanticipated (Serious) Adverse Device Effect (UADE), the Investigator will submit a report of the UADE to the Sponsor and IEC/IRB as soon as possible, but no later than 24 hours after the Investigator first learns of the effect. This report is in addition to the immediate notification mentioned above.

The Sponsor must conduct an evaluation of the UADE and must report the results of the evaluation to FDA, the IEC/IRB and participating Investigators within 10 working days after the Sponsor first receives notification of the effect.

#### **Non-Serious Adverse Events**

All non-serious adverse events, including non-serious adverse device effects, will be reported to the sponsor by the Investigator no later than 2 days from discovery.

# 13.4.2. Reporting Adverse Events to the Responsible IEC/IRB and Health Authorities

Adverse events that meet the IEC/IRB requirements for reporting must be reported within the IEC/IRB's written guidelines. Each clinical site will refer to and follow any guidelines set forth by their Approving IEC/IRB. Each clinical site will refer to and follow any guidelines set forth by their local governing Health Authorities.

The Sponsor will report applicable Adverse Events to the local health authorities according the written guidelines, including reporting timelines.

# 13.4.3. Event of Special Interest

None.

# 13.5. Reporting of Pregnancy

Subjects reporting pregnancy (by self-report) during the study will be discontinued after the event is recorded as an Adverse Event. Once discontinued, pregnant participants and their fetuses will not be monitored for study related purposes. At the Investigator's discretion, the study participant may be followed by the Investigator through delivery. However, this data will not be collected as part of the clinical study database. Pregnant participants are not discontinued from contact lens or solution related studies for safety concerns, but due to general concerns relating to pregnancy and contact lens use. Specifically, pregnant women are discontinued due to fluctuations in refractive error and/or visual acuity that occur secondary to systemic hormonal changes, and not due to unforeseen health risks to the mother or fetus.

#### 14. STATISTICAL METHODS

#### 14.1. General Considerations

All data summaries and statistical analyses will be performed using the SAS software Version 9.4 or higher (SAS Institute, Cary, NC). Throughout the analysis of data, the results for each subject/eye will be used when available for summarization and statistical analysis. Unscheduled visits will be summarized separately and will be excluded from the statistical analysis.

Summary tables (Descriptive statistics and/or frequency tables) will be provided for all baseline variables, efficacy variables and safety variables as appropriate. Continuous variables will be summarized with descriptive statistics (n, mean, standard deviation (SD), median, minimum and maximum). Frequency count and percentage of subjects or eyes within each category will be provided for categorical data.

Summaries will be presented by study lens type and will be performed separately by completion status. All analyses will be conducted on per-protocol population (see Section 14.3).

# 14.2. Sample Size Justification

A total of approximately 40 eligible subjects will be enrolled into the study at this site. At least 36 subjects will complete this study.

Using the POWER procedure in SAS 9.4, below is the summary of sample size required based on the different assumptions of the true LogMAR visual acuity and CLUE scores. The sample size was calculated for the non-inferiority tests (using 0.05 as the margin) with at least 90% of statistical power and 2-sided type I error of 0.05. Assuming the true LogMAR visual acuity is between 0.00 to 0.05 (distance) or 0.08 to 0.12 (near), and true CLUE vision score is between 38 to 42 points.

# • Binocular LogMAR visual acuity (distance)

| | Estimated Standard | | Actual |
|------------|--------------------|----------------------|--------|
| True Value | Deviation | # of subjects needed | Power |
| 0.00 | 0.12 | 18 | 0.915 |
| 0.02 | 0.12 | 26 | 0.904 |
| 0.05 | 0.12 | 63 | 0.902 |

#### • Binocular LogMAR visual acuity (near)

| | Estimated Standard | | Actual |
|------------|--------------------|----------------------|--------|
| True Value | Deviation | # of subjects needed | Power |
| 0.08 | 0.12 | 21 | 0.905 |
| 0.10 | 0.12 | 33 | 0.901 |
| 0.12 | 0.12 | 63 | 0.902 |

# • CLUE vision score

| | Estimated Standard | | Actual |
|------------|--------------------|----------------------|--------|
| True Value | Deviation | # of subjects needed | Power |
| 38 | 17 | 87 | 0.902 |
| 40 | 17 | 50 | 0.903 |
| 42 | 17 | 33 | 0.906 |

# 14.3. Analysis Populations

# **Safety Population:**

All subjects who were administered any test article excluding subjects who drop out prior to administering any test article. At least one observation should be recorded.

## **Per-Protocol Population:**

All subjects who have successfully completed all visits and did not substantially deviate from the protocol as determined by the trial cohort review committee prior to database hard lock (Per-Protocol Population). Justification of excluding subjects with protocol deviations in the per-protocol population set will be documented in a memo to file.

# **Intent-to-Treat (ITT) Population:**

All assigned subjects regardless of actual treatment and subsequent withdrawal from study or deviation from protocol. At least one observation should be recorded.

# 14.4. Level of Statistical Significance

All planned analysis for this study will be conducted with an overall type I error rate of 5%.

# 14.5. Primary Analysis

# **LogMAR Visual Acuity**

Binocular, high luminance, high contrast visual performance on logMAR scale will be analyzed using a linear mixed model. Each regression model will include the experimental design factors: distance as fixed effects. Other baseline characteristics known of importance such as age, gender, and/or add power will be included as fixed covariates when appropriate. Subject nested in site will be included as random covariates when appropriate. The covariance between residual errors from the same subject across different charts will be selected based on the finite-sample corrected Akaike's Information Criterion.<sup>6</sup> Covariance structures considered may include: Homogenous compound symmetry (CS) and Unstructured covariance structure (UN). The structure that returns the lowest Akaike Information Criteria Corrected (AICC) will be selected as the structure that best fit the data.

Comparisons will be carried out using 95% confidence intervals constructed of least-square means (LSM) from the linear mixed models. Statistically superiority will be concluded if the upper limits of the confidence intervals are below the thresholds for corresponding distances.

# **CLUE Vision Scores**

CLUE vision scores will be analyzed using a linear mixed model adjusting for baseline values as fixed covariate. The model will include the experimental design factors: time (6-8 day or 12-16 day) as fixed effects. Other baseline characteristics known of importance such as age, gender, and/or add power will be included as fixed covariates when appropriate. The covariance between residual errors from the same subject across different time will be selected based on the finite-sample corrected Akaike's Information Criterion. Covariance structures considered may include: Homogenous compound symmetry (CS) and Unstructured covariance structure (UN). The structure that returns the lowest Akaike Information Criteria Corrected (AICC) will be selected as the structure that best fit the data.

Comparisons will be carried out using 95% confidence intervals constructed of least-square means (LSM) from the linear mixed models for each time. Statistically superiority will be concluded if the lower limit of the confidence interval is greater than 32 points.

In all models, the Kenward and Roger method<sup>7</sup> will be used for the calculation of the denominator of degrees of freedom.

# 14.6. Secondary Analysis

Not Applicable.

## 14.7. Other Exploratory Analyses

Not Applicable.

## 14.8. Interim Analysis

Not Applicable.

# 14.9. Procedure for Handling Missing Data and Drop-Outs

Missing or spurious values will not be imputed. The count of missing values will be included in the summary tables and listings.

Subject dropout is expected to be one of the main reasons of missing data in this clinical trial. Past clinical trials don't provide the evidence that subject dropout is systematic or not-at-random. To evaluate the impact of missing data, sensitivity analysis will be conducted using multiple imputation methods if the proportion of subject dropout is greater than the 15%. The SAS/STAT procedures PROC MI and PROC MIANALYZE will be utilized with a parametric regression method used to make at least 5 imputations.

#### 14.10. Procedure for Reporting Deviations from Statistical Plan

The analysis will be conducted according to that specified in above sections. There are no known reasons for which it is planned to deviate from these analysis methods. If for any reason a change is made, the change will be documented in the study report along with a justification for the change.

#### 15. DATA HANDLING AND RECORD KEEPING/ARCHIVING

# 15.1. Electronic Case Report Form/Data Collection

The data for this study will be captured on electronic case report forms (eCRFs) using an EDC system (Bioclinica). An authorized data originator will enter study data into the eCRFs using the EDC system. Data collected on equipment that is not captured in EDC will be formatted to the specification of the JJVC database manager and sent to JJVC for analysis

The clinical data will be recorded on dedicated eCRFs specifically designed to match the study procedures for each visit. Once completed, the eCRFs will be reviewed for accuracy and completeness and signed by the Investigator. The sponsor or sponsor's representatives will be authorized to gain access to the subject recordation for the purposes of monitoring and auditing the study.

Edit checks, electronic queries, and audit trails are built into the system to ensure accurate and complete data collection. Data will be transmitted from the clinical site to a secure central database as forms are completed or updated, ensuring information accuracy, security, and confidentiality. After the final database lock, the Investigator will be provided with Individual Patient Profiles (IPP) including the full audit trail on electronic media in PDF format for all of the study data. The IPP must be retained in the study files as a certified copy of the source data for the study.

The content and structure of the eCRFs are compliant with ISO14155:2011.<sup>1</sup>

# 15.2. Subject Record

At a minimum, subject record should be available for the following:

- subject identification
- eligibility
- study identification
- study discussion
- provision of and date of informed consent
- visit dates
- results of safety and efficacy parameters as required by the protocol
- a record of all adverse events
- follow-up of adverse events
- medical history and concomitant medication
- test article receipt/dispensing/return records
- date of study completion
- reason for early discontinuation of test article or withdrawal from the study, if applicable

The subject record is the eCRF or an external record. The author of an entry in the subject record must be identifiable. The first point of entry is considered to be the source record.

Adverse event notes must be reviewed and initialed by the Investigator.

#### 16. DATA MANAGEMENT

#### 16.1. Access to Source Data/Document

The Investigator/Institution will permit trial-related monitoring, audits, IEC/IRB review and regulatory inspection(s) by providing direct access to source data/documents. Should the clinical site be contacted for an audit by an IEC/IRB or regulatory authority, JJVC must be contacted and notified in writing within 24 hours.

## 16.2. Confidentiality of Information

Information concerning the investigational product and patent application processes, scientific data or other pertinent information is confidential and remains the property of JJVC. The Investigator may use this information for the purposes of the study only. It is understood by the Investigator that JJVC will use information developed in this clinical study in connection with the development of the investigational product and therefore may disclose it as required to other clinical investigators and to regulatory agencies. In order to allow the use of the information derived from this clinical study, the Investigator understands that he/she has an obligation to provide complete test results and all data developed during this study to the Sponsor.

## 16.3. Data Quality Assurance

Steps will be taken to ensure the accuracy and reliability of data, include the selection of qualified investigators and appropriate clinical sites and review of protocol procedures with the Principal Investigator. The Principal Investigator, in turn, must ensure that all Sub-Investigators and clinical site personnel are familiar with the protocol and all study-specific procedures and have appropriate knowledge of the study article.

Training on case report form completion will be provided to clinical site personnel before the start of the study. The Sponsor will review case report forms for accuracy and completeness remotely during the conduct of the study, during monitoring visits, and after transmission to data management. Any data discrepancies will be resolved with the Investigator or designee, as appropriate.

Quality Assurance representatives from JJVC may visit clinical sites to review data produced during the study and to access compliance with applicable regulations pertaining to the conduct of clinical trials. The clinical sites will provide direct access to study-related source data/documents and reports for the purpose of monitoring and auditing by JJVC and for inspection by local and regulatory authorities.

#### 17. MONITORING

The study monitors will maintain close contact with the Principal Investigator and the Investigator's designated clinical site personnel. The monitor's responsibilities will include:

- Ensuring that the investigation is being conducted according to the protocol, any subsequent amendments, and regulatory requirements are maintained
- Ensuring the rights and wellbeing of subjects are protected
- Ensuring adequate resources, including facilities, laboratories, equipment, and qualified clinical site personnel
- Ensuring that protocol deviations are documented with corrective action plans, as applicable
- Ensuring that the clinical site has sufficient test article and supplies
- Clarifying questions regarding the study
- Resolving study issues or problems that may arise
- Reviewing of study records and source documentation verification in accordance with the monitoring plan

#### 18. ETHICAL AND REGULATORY ASPECTS

## 18.1. Study-Specific Design Considerations

Potential subjects will be fully informed of the risks and requirements of the study and, during the study, subjects will be given any new information that may affect their decision to continue participation. Subjects will be told that their consent to participate in the study is voluntary and may be withdrawn at any time with no reason given and without penalty or loss of benefits to which they would otherwise be entitled. Only subjects who are fully able to understand the risks, benefits, and potential adverse events of the study, and provide their consent voluntarily will be enrolled.

## 18.2. Investigator Responsibility

The Principal Investigator is responsible for ensuring that the clinical study is performed in accordance with the signed agreement, the investigational plan, Section 4 of the ICH E6 guidelines on Good Clinical Practice (GCP),<sup>2</sup> and applicable regulatory requirements. GCP is an international ethical and scientific quality standard for designing, conducting, recording, and reporting studies that involve the participation of human subjects. Compliance with this standard provides public assurance that the rights, safety, and well-being of study subjects are protected, consistent with the principles of the Declaration of Helsinki 64<sup>th</sup> WMA General Assembly 2013<sup>3</sup> and that the clinical study data are credible. The Investigator must maintain clinical study files in accordance with Section 8 of the ICH E6 guidelines on Good Clinical Practice (GCP),<sup>2</sup> and applicable regulatory requirements.

# 18.3. Independent Ethics Committee or Institutional Review Board (IEC/IRB)

Before the start of the study, the Investigator (or Sponsor when applicable) will provide the IEC/IRB with current and complete copies of the following documents (where applicable):

- Final protocol and, if applicable, amendments
- Sponsor-approved informed consent form (and any other written materials to be provided to the subjects)
- Investigator's Brochure (or equivalent information) and amendments
- Sponsor-approved subject recruitment materials
- Information on compensation for study-related injuries or payment to subjects for participation in the study
- Investigator's curriculum vitae, clinical licenses, or equivalent information (unless not required, as documented by IEC/IRB)
- Information regarding funding, name of the Sponsor, institutional affiliations, other potential conflicts of interest, and incentives for subjects
- Any other documents that the IEC/IRB requests to fulfill its obligation

This study will be undertaken only after IEC/IRB has given full approval of the final protocol, amendments (if any), the informed consent form, applicable recruiting materials, and subject compensation programs, and the Sponsor has received a copy of this approval. This approval letter must be dated and must clearly identify the documents being approved.

During the study, the Investigator (or Sponsor when applicable) will send the following documents to the IEC/IRB for their review and approval, where appropriate:

- Protocol amendments
- Revision(s) to informed consent form and any other written materials to be provided to subjects
- If applicable, new or revised subject recruitment materials approved by the Sponsor
- Revisions to compensation for study-related injuries or payment to subjects for participation in the study
- Investigator's Brochure amendments or new edition(s)
- Summaries of the status of the study (at least annually or at intervals stipulated in guidelines of the IEC/IRB)
- Reports of adverse events that are serious, unanticipated, and associated with the test articles, according to the IRB's requirements
- New information that may adversely affect the safety of the subjects or the conduct of the study
- Major protocol deviations as required by the IEC/IRB
- Report of deaths of subjects under the Investigator's care
- Notification if a new Investigator is responsible for the study at the clinical site
- Any other requirements of the IEC/IRB

For protocol amendments that increase subject risk, the amendment and applicable informed consent form revisions must be submitted promptly to the IEC/IRB for review and approval before implementation of the change(s).

At least once a year, the IEC/IRB will review and reapprove this clinical study. This request should be documented in writing.

At the end of the study, the Investigator (or Sponsor where required) will notify the IEC/IRB about the study completion. Documentation of this notification must be retained at the clinical site and a copy provided to the CRO or Sponsor as applicable.

## 18.4. Informed Consent

Each subject must give written consent according to local requirements after the nature of the study has been fully explained. The consent form must be signed before performance of any study-related activity. The consent form that is used must be approved by both the Sponsor and by the reviewing IEC/IRB. The informed consent is in accordance with principles that originated in the Declaration of Helsinki,<sup>3</sup> current ICH<sup>2</sup> and ISO 14155<sup>1</sup> guidelines, applicable regulatory requirements, and Sponsor Policy.

Before entry into the study, the Investigator or an authorized member of the clinical site personnel must explain to potential subject the aims, methods, reasonably anticipated benefits, and potential hazards of the study, and any discomfort it may entail. Subjects will be informed that their participation is voluntary and that they may withdraw consent to participate at any time.

The subject will be given sufficient time to read the informed consent form and the opportunity to ask questions. After this explanation and before entry into the study, consent should be appropriately recorded by means of the subject's dated signature. After having obtained the consent, a copy of the informed consent form must be given to the subject.

## 18.5. Privacy of Personal Data

The collection, processing and disclosure of personal data and medical information related to the Study Subject, and personal data related to Principal Investigator and any clinical site personnel (e.g., name, clinic address and phone number, curriculum vitae) is subject to compliance with the Health Information Portability and Accountability Act (HIPAA) in the United States<sup>4</sup> and other applicable personal data protection and security laws and regulations. Appropriate measures will be employed to safeguard these data, to maintain the confidentiality of the person's related health and medical information, to properly inform the concerned persons about the collection and processing of their personal data, to grant them reasonable access to their personal data and to prevent access by unauthorized persons.

All information obtained during the course of the investigation will be regarded as confidential. All personal data gathered in this trial will be treated in strictest confidence by Investigators, monitors, Sponsor's personnel and IEC/IRB. No data will be disclosed to any third party without the express permission of the subject concerned, with the exception of Sponsor personnel (monitor, auditor), IEC/IRB and regulatory organizations in the context of their investigation related activities that, as part of the investigation will have access to the CRFs and subject records.

The collection and processing of personal data from subjects enrolled in this study will be limited to those data that are necessary to investigate the efficacy, safety, quality, and utility of the investigational product(s) used in this study.

These data must be collected and processed with adequate precautions to ensure confidentiality and compliance with applicable data privacy protection laws and regulations.

The Sponsor ensures that the personal data will be:

- processed fairly and lawfully
- collected for specified, explicit, and legitimate purposes and not further processed in a way incompatible with these purposes
- adequate, relevant, and not excessive in relation to said purposes
- accurate and, where necessary, kept current

Explicit consent for the processing of personal data will be obtained from the participating subject before collection of data. Such consent should also address the transfer of the data to other entities and to other countries.

The subject has the right to request through the Investigator access to his personal data and the right to request rectification of any data that are not correct or complete. Reasonable steps should be taken to respond to such a request, taking into consideration the nature of the request, the conditions of the study, and the applicable laws and regulations.

Appropriate technical and organizational measures to protect the personal data against unauthorized disclosures or access, accidental or unlawful destruction, or accidental loss or alteration must be put in place. Sponsor personnel whose responsibilities require access to personal data agree to keep the identity of study subjects confidential.

#### 19. STUDY RECORD RETENTION

In compliance with the ICH/GCP guidelines,<sup>2</sup> the Investigator/Institution will maintain all CRFs and all subject records that support the data collected from each subject, as well as all study documents as specified in ICH/GCP<sup>2</sup> and all study documents as specified by the applicable regulatory requirement(s). The Investigator/Institution will take measures to prevent accidental or premature destruction of these documents.

Essential documents must be retained until at least two (2) years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated marketing applications in an ICH region or until at least two (2) years have elapsed since the formal discontinuation of clinical development of the investigational product. These documents will be retained for a longer period if required by the applicable regulatory requirements or instructed by the Sponsor. It is the responsibility of the Sponsor to inform the Investigator/Institution as to when these documents no longer need to be retained.

If the responsible Investigator retires, relocates, or for other reasons withdraws from the responsibility of keeping the study records, custody must be transferred to a person who will accept the responsibility. The Sponsor must be notified in writing of the name and address of the new custodian. Under no circumstance shall the Investigator relocate or dispose of any study documents before having obtained written approval from the Sponsor.

If it becomes necessary for the Sponsor or the appropriate regulatory authority to review any documentation relating to this study, the Investigator must permit access to such reports. If the Investigator has a question regarding retention of study records, he/she should contact JJVC.

#### 20. FINANCIAL CONSIDERATIONS

Remuneration for study services and expenses will be set forth in detail in the Clinical Research Agreement. The Research Agreement will be signed by the Principal Investigator and a JJVC management representative prior to study initiation.

JJVC reserves the right to withhold remuneration for costs associated with protocol violations such as:

- Continuing an ineligible subject in the study
- Scheduling a study visit outside the subject's acceptable visit range

JJVC reserves the right to withhold final remuneration until all study related activities have been completed, such as:

- Query resolution
- Case Report Form signature
- Completion of any follow-up action items

#### 21. PUBLICATION

This study will be registered on ClinicalTrials.gov by the Sponsor.

#### 22. REFERENCES

- 1. ISO 14155:2011: Clinical Investigation of Medical Devices for Human Subjects Good Clinical Practice. Available at: <a href="https://www.iso.org/standard/45557.html">https://www.iso.org/standard/45557.html</a>
- 2. International Conference on Harmonization Good Clinical Practice E6 (ICH-GCP). Available at: <a href="http://www.ich.org/products/guidelines/efficacy/article/efficacy-guidelines.html">http://www.ich.org/products/guidelines/efficacy/article/efficacy-guidelines.html</a>
- 3. Declaration of Helsinki Ethical principles for Medical Research Involving Human Subjects. Available at: <a href="https://www.wma.net/policies-post/wma-declaration-of-helsinki-ethical-principles-for-medical-research-involving-human-subjects/">https://www.wma.net/policies-post/wma-declaration-of-helsinki-ethical-principles-for-medical-research-involving-human-subjects/</a>
- 4. United States (US) Code of Federal Regulations (CFR). Available at: <a href="https://www.gpo.gov/fdsys/browse/collectionCfr.action?collectionCode=CFR">https://www.gpo.gov/fdsys/browse/collectionCfr.action?collectionCode=CFR</a>
- 5. Health Information Portability and Accountability Act (HIPAA). Available at: <a href="https://www.hhs.gov/hipaa/for-professionals/privacy/index.html">https://www.hhs.gov/hipaa/for-professionals/privacy/index.html</a>
- 6. Keselman HJA, J.; Kowalchuk, R. K.; and Wolfinger, R. D. A Comparison of Two Approaches for Selecting Covariance Structures in the Analysis of Repeated Measures. *Communications in Statistics—Simulation and Computation*. 1998;27(3):591–604.
- 7. Kenward MG and Roger JH. Small Sample Inference for Fixed Effects from Restricted Maximum Likelihood. *Biometrics*, 1997;53:983–997.

# APPENDIX A: PATIENT REPORTED OUTCOMES (STUDY QUESTIONNAIRES)






CR-6278, v1.0 JJVC Confidential PRO SPECIFICATION Version 1 Final 2018-06-13 
6

CR-6278, v1.0


CR-6278, v1.0


CR-6278, v1.0 JJVC Confidential PRO SPECIFICATION Version 1 Final 2018-06-13 

CR-6278, v1.0



CR-6278, v1.0





CR-6278, v1.0 JJVC Confidential PRO SPECIFICATION Version 1 Final 2018-06-13

16

## APPENDIX B: PATIENT INSTRUCTION GUIDE

# APPENDIX C: PACKAGE INSERT (APPROVED PRODUCT)

Not Applicable

#### APPENDIX D: PRESBYOPIC SYMPTOMS QUESTIONNAIRE



#### APPENDIX E: OCULAR DOMINANCE



## APPENDIX F: TEST LENS FITTING GUIDE





#### APPENDIX G: BINOCULAR OVER REFRACTION



#### **APPENDIX H:**

- LIMBAL & CONJUNCTIVAL (BULBAR) REDNESS
- EXPANDED SODIUM FLUORESCEIN CORNEAL STAINING
- DETERMINATION OF NEAR ADD
- NEAR logMAR VISUAL ACUITY MEASUREMENT PROCEDURE
- LENS FITTING CHARACTERISTICS
- SUBJECT REPORTED OCULAR SYMPTOMS
- DETERMINATION OF DISTANCE SPHEROCYLINDRICAL REFRACTIONS
- BIOMICROSCOPY SCALE
- KERATOMETRY
- DISTANCE AND NEAR VISUAL ACUITY EVALUATION
- TORIC FIT EVALUATION
- ETDRS DISTANCE VISUAL ACUITY MEASURMENT PROCEDURE
- LENS INSERTION AND REMOVAL
- VISUAL ACUITY CHART LUMINANCE AND ROOM ILLUMINATION
  TESTING

## LIMBAL & CONJUNCTIVAL (BULBAR) REDNESS






JJVC Confidential











# EXPANDED SODIUM FLUORESCEIN CORNEAL STAINING










## **DETERMINATION OF NEAR ADD**

















#### NEAR LOGMAR VISUAL ACUITY MEASUREMENT PROCEDURE






### LENS FITTING CHARACTERISTICS














## SUBJECT REPORTED OCULAR SYMPTOMS



# DETERMINATION OF DISTANCE SPHEROCYLINDRICAL REFRACTIONS


















### BIOMICROSCOPY SCALE











JJVC Confidential


CR-6278, v1.0



### KERATOMETRY



## DISTANCE AND NEAR VISUAL ACUITY EVALUATION


| Distance and Near Visual Acuity Evaluation | |
|--------------------------------------------|--------------------|
| Clinical Test Procedure | |
| | Revision Number: 3 |
| * | |

| Title: | Distance and Near Visual Acuity Evaluation | |
|---|---|---|
| <b>Document Type:</b> | Clinical Test Procedure | |
| Document Number: | | Revision Number: 3 |
## TORIC FIT EVALUATION








#### ETDRS DISTANCE VISUAL ACUITY MEASURMENT PROCEDURE

| Title: | Distance LogMAR Visual Acuity Measurement Procedure | |
|---|---|---|
| <b>Document Type:</b> | <b>Clinical Test Procedure</b> | |
| Document Number: | | Revision Number: 4 |




## LENS INSERTION AND REMOVAL

Title: Lens Insertion and Removal

Document Type: Work Instructions

Document Number: Revision Number: 2

# VISUAL ACUITY CHART LUMINANCE AND ROOM ILLUMINATION TESTING






**Visual Acuity Chart Luminance and Room Illumination Testing** 

Title:

#### PROTOCOL COMPLIANCE INVESTIGATOR(S) SIGNATURE PAGE

Protocol Number and Title: CR-6278 Evaluation of a Toric Multifocal Contact Lens Manufactured in Etafilcon Material in a Low ADD Hyperopic Population

Version and Date: 1.0 12 July 2018

I have read and understand the protocol specified above and agree on its content.

I agree to conduct this study according to ISO 14155,<sup>1</sup> GCP and ICH guidelines,<sup>2</sup> the Declaration of Helsinki,<sup>3</sup> United States (US) Code of Federal Regulations (CFR),<sup>4</sup> and the pertinent individual country laws/regulations and to comply with its obligations, subject to ethical and safety considerations. The Principal Investigator is responsible for ensuring that all clinical site personnel, including Sub-Investigators adhere to all ICH<sup>2</sup> regulations and GCP guidelines regarding clinical trials during and after study completion.

I will assure that no deviation from, or changes to the protocol will take place without prior agreement from the Sponsor and documented approval from the Institutional Review Board (IRB), except where necessary to eliminate an immediate hazard(s) to the trial participants.

I am responsible for ensuring that all clinical site personnel including Sub-Investigators adhere to all ICH<sup>2</sup> regulations and GCP guidelines regarding clinical trials during and after study completion.

All clinical site personnel involved in the conduct of this study have completed Human Subjects Protection Training.

I agree to ensure that all clinical site personnel involved in the conduct of this study are informed about their obligations in meeting the above commitments.

I shall not disclose the information contained in this protocol or any results obtained from this study without written authorization.

| Principal Investigator: | | |
|-------------------------|------------------------------------------|------|
| | Signature | Date |
| | Name and Professional Position (Printed) | - |
| Institution/Site: | | |
| | Institution/Site Name | |
| | Institution/Site Address | |